Project ID: IIR 19-013, eRA# 101 HX003060-01

Funding Agency: VA HSR&D

Principal Investigator/Study Chair: Deborah Gurewich, PhD

Version: 11/06/2023


#### Abstract

**Background:** Despite medical advances, up to 70% of health outcomes are due to social determinants of health (SDoH) - the conditions in which people live and work that shape whether basic needs (e.g., housing, food) are met. These associations are especially well documented for cardiovascular disease (CVD). In response, health policy leaders recommend screening and referral (S&R) for unmet needs in clinical settings, and the American Heart Association recently concluded that the most significant opportunities for reducing CVD death and disability lie with addressing the social determinants of cardiovascular outcomes. A limited but promising evidence base supports these recommendations, but more rigorous research is needed to guide how best to intervene on unmet needs that affect health.

Innovation: VA currently systematically screens for only two unmet needs (homelessness and food insecurity). Identification of other unmet needs (and referral to address them) occurs on an ad hoc basis, with varying approaches among clinics/ clinicians. We will implement comprehensive screening of nine unmet needs and systematic referral, developing tools and processes that, if efficacious, can be implemented within VA (and other) clinical systems. VA is currently funding several studies related to SDoH, but none test interventions that systematically identify a wide range of unmet social needs among Veterans and connect Veterans with identified needs to social service resources.

Specific Aims: 1) Describe the burden and distribution of nine unmet needs (i.e., housing; food insecurity; utility insecurity; transportation; legal guidance; employment; safety; and social isolation) among Veterans with or at-risk for CVD, and identify their associations with sociodemographic characteristics, and baseline health-related behaviors and clinical outcomes; 2) Compare the effects of three S&R study intervention conditions of varying intensity on Veterans' connection to new SDoH resources (primary outcome), reduction of unmet needs, adherence, and clinical outcomes, and 3) Identify barriers and facilitators to Veterans' connecting with social services and having needs met, and explanatory factors for observed RCT outcomes.

Methodology: We propose a three-year, two-phased mixed methods study. In Phase One (Aims 1 and 2), we will implement a three-armed randomized controlled trial at three VA sites to compare outcomes among Veterans randomized within each site to one of three study conditions: screening only; screening plus provision of tailored resource sheets; or screening plus resource sheets plus social work support. For each Veteran, we will examine associations


of unmet needs with baseline outcomes (Aim 1), and longitudinally examine the impact of each approach on connection to new SDoH resources and follow-up outcomes over a 12-month period (Aim 2). In Phase Two (Aim 3), we will conduct interviews with Veterans and representatives of the VA- and community-based programs to which Veterans are referred because of the trial to identify facilitators and barriers and potential explanatory factors related to the relative success of the interventions.


3

VA Central IRB Effective Date: November 29, 2023

#### List of Abbreviations

ACO Accountable Care Organization

ACSC Ambulatory Care Sensitive Conditions

AHA American Heart Association

AHC Accountable Health Communities

AHRQ Agency for Healthcare Research and Quality

**BMC Boston Medical Center** 

**BP Blood Pressure** 

BS Bachelor of Science

CDC Centers for Disease Control and Prevention

CDW Corporate Data Warehouse

CHC Community Health Center

CHERP Center for Health Equity Research and Promotion

CHF Congestive Heart Failure

CHOIR Center for Healthcare Organization and Implementation Research

CMS Center for Medicare and Medicaid Services

CPT Current Procedure Terminology

CVD Cardiovascular Disease

**ED Emergency Department** 

EHR Electronic Health Record

HbA1c Hemoglobin A1c

HSR&D Health Services Research and Development

4

ICD10 International Classification of Disease 10th Revision

IIR Investigator-Initiated Research

IOM Institutes of Medicine

MLCHC Massachusetts League of Community Health Centers

MPH Master of Public Health

MPI Multiple Principal Investigators

MSW Master of Social Work

NACHC National Association of Community Health Centers

NAM National Academy of Medicine

NHLBI National Heart, Lung and Blood Institute

NIH National Institutes of Health

OPCC&CT Office of Patient Centered Care & Cultural Transformation

PC Primary Care

PI Principal Investigator

**PQI Preventative Quality Indicators** 

PRAPARE Protocol for Patients' Assets, Risk, and Experiences

RA Research Associate

S&R Screening and Referring

SDoH Social Determinants of Health

**SEP Socioeconomic Position** 

VACS Veteran Aging Cohort Study

VERG Veterans Employee Resource Group

VINCI VA Informatics and Computing Infrastructure

5

VIReC VA Information Resource Center

VISTA Veterans Health Information Systems and Technology Architecture

VSSC VHA Support Service Center

WHO World Health Organization

# **Contents**

| | ocol Title: The Effects of Screening and Referral for Social Determinants | |
|---|---|---|
| on V | /eterans' Outcomes | 8 |
| 1.0 | Study Personnel | 8 |
| 2.0 | Introduction | 8 |
| 3.0 | Objectives | 10 |
| 4.0 | Resources and Personnel | 11 |
| 5.0 | Study Procedures | 15 |
| 5. | 1 Study Design | 15 |
| 5. | 2 Recruitment Methods | 21 |
| 5. | 3 Informed Consent Procedures | 24 |
| 5. | 4 Inclusion/Exclusion Criteria | 24 |
| 5. | 5 Study Evaluations | 25 |
| 5. | 6 Data Analysis | 26 |
| 5. | 7 Withdrawal of Subjects | 31 |
| 6.0 | Reporting | 31 |
| 7.0 | Privacy and Confidentiality | 31 |
| 8.0 | Communication Plan | 32 |
| 9.0 | References | 32 |
| Αŗ | ppendix A: Description of the Intervention and Randomization | 34 |
| Αŗ | ppendix B: Protocol for Warm Hand-Off to Veterans Crisis Line | 37 |
| Αŗ | ppendix C: Cover Letter Inviting Veteran Participation | 40 |
| Αŗ | ppendix D: Study Fact Sheet | 41 |
| Αŗ | ppendix E: Sample Resource Postcards | 44 |
| Αŗ | ppendix F: Opt-Out (Do-not-contact) Postcard | 44 |
| Αŗ | ppendix G: Veteran Recruitment Phone Script | 46 |
| Αŗ | ppendix H: Resource Representative Invitation Email | 54 |
| Αp | ppendix I: Index Unmet Needs Screening Tool | 54 |
| Αp | ppendix J: Eight-Week Follow-Up Survey | 59 |
| Αŗ | ppendix K: Six-Month Follow-Up Survey | 61 |

| Appendix L: Veteran Interview Guide (Not Connected) | 64 |
|---|---|
| Appendix M: Veteran Interview Guide (Connected) | 67 |
| Appendix N: Resource Representative Interview Guide | 70 |
| Appendix O: Example Resource Sheets | 72 |
| Appendix P. Mail and Email Text for Delivering Resource Sheets to Veterans | 81 |

# Protocol Title: The Effects of Screening and Referral for Social Determinants of Health on Veterans' Outcomes

# 1.0 Study Personnel

| Name | Project<br>Role | Status | Email | Institution and Location |
|---|---|---|---|---|
| Gurewich, | PI | 8/8ths | Deborah.Gurewich@va.gov | VA Boston Healthcare |
| Deborah | | VA | | System, Boston, MA |
| Rosen, Amy | co-l | 8/8ths<br>VA | Amy.Rosen2@va.gov | VA Boston Healthcare<br>System, Boston, MA |
| Niles, Barbara | co-l | 8/8ths<br>VA | Barbara.Niles@va.gov | VA Boston Healthcare<br>System, Boston, MA |
| Linsky, Amy | co-l | 8/8ths<br>VA | Amy.Linsky@va.gov | VA Boston Healthcare<br>System, Boston, MA |
| Friedman,<br>Hannah | Co-I | 8/8ths<br>VA | Hannah.Friedman2@va.gov | VA Boston Healthcare<br>System, Boston, MA |
| Bokhour,<br>Barbara | co-l | 8/8ths<br>VA | Barbara.Bokhour@va.gov | Edith Nourse Rogers<br>Memorial Veterans<br>Hospital (Bedford VAMC),<br>Bedford, MA |
| Fix, Gemmae | co-l | 8/8ths<br>VA | Gemmae.Fix@va.gov | Bedford VAMC, Bedford,<br>MA |
| Li, Mingfei | co-l | IPA | Mingfei.Li@va.gov | Bedford VAMC, Bedford, MA |
| Hunt, Kelly | co-l | 8/8ths<br>VA | Kelly.Hunt@va.gov | Ralph H Johnson Medical<br>Center, Charleston, MA |
| Dichter, Melissa | co-l | 8/8ths<br>VA | Melissa.Dichter@va.gov | Corporal MJ Crescenz VA<br>Medical Center,<br>Philadelphia, PA |

Four sites will participate in this study, 3 of which are intervention sites
(Boston, Charleston and Philadelphia) and 1 of which is a non-intervention
site (Bedford). Team members at the non-intervention site will only be
engaged in advising the study, qualitative data analysis, and
dissemination activities. There is not a graduated start-up plan for any of
the sites.

## 2.0 Introduction

8

Credit for health outcomes is typically ascribed to biomedical advances, but up to 70% of health outcomes result from social determinants of health (SDoH) -- the conditions in which individuals are born, live and work. SDoH shape whether basic needs (e.g., housing, utilities, food, transportation, employment, social connections, legal assistance, safety) are met.<sup>1, 2</sup> As posited by Maslow's hierarchy of needs model,<sup>3</sup> individuals' **unmet needs** can affect adherence to medical therapies and outpatient care appointments, preventable hospitalizations and urgent care use, and ultimately, health outcomes. These associations are well documented for cardiovascular disease (CVD), the leading cause of morbidity and mortality in the US. <sup>4-6</sup> Given the simultaneously high prevalence of CVD and its risk factors and unmet needs among Veterans, Veterans' outcomes may be improved by comprehensively assessing and addressing unmet needs. <sup>7</sup>

In fact, policymakers suggest routine, comprehensive screening for unmet needs in the clinical setting. <sup>8</sup> The American Heart Association recently concluded that the "most significant opportunities for reducing CVD death and disability lie with addressing the social determinants of CVD outcomes." <sup>9</sup> These recommendations rest on limited, yet promising, evidence that implementing systematic screening and referral (S&R) for unmet needs leads to greater receipt of resources that address identified needs. <sup>10, 11</sup> Such a process can potentially improve both proximal outcomes, such as adherence to medications and care appointments, <sup>12</sup> as well as more distal outcomes, such as inpatient or urgent health care utilization and ideally, overall improved health. <sup>13-15</sup>

Currently, the VA has implemented nationwide, clinic-based S&R for two unmet needs (housing and food insecurity) and invests in social work (SW) to address a range of unmet needs. VA clinicians can refer patients to SW to address unmet needs; patients may also self-refer. Once connected to SW, Veterans are triaged, a bio-psychosocial assessment identifies unmet needs, and SWs facilitate referrals to resources to assist with identified needs. However, and of crucial importance, screening for a wider range of unmet needs (beyond housing and food) and referring to SW is ad hoc and highly variable across and within facilities. Thus, many Veterans who could benefit from VA SW are not systematically identified and referred.

VAs' lack of systematic and comprehensive S&R for unmet needs also means missed opportunities to better understand the scope and scale of unmet needs across the entire VA patient population, as no such data exists. <sup>14</sup> This in turn limits VA's understanding of how best to support and target SW services. It is also unknown whether a lower-intensity referral process (i.e., provision of tailored paper Resource Sheets to address unmet needs instead of a referral to SW) can help some Veterans to the same extent it helps patients in non-VA care settings.

<sup>10, 16</sup> Thus, a critically important dimension of the study we propose is to test whether for some Veterans, a less intense intervention is adequate. If so, this has valuable implications for resource allocation decisions and future implementation.

To address these knowledge gaps, we propose a **randomized controlled trial** (RCT) to systematically screen Veterans with/at risk for CVD for nine unmet needs, characterize the prevalence of unmet needs and associations with outcomes, and compare the effect of two different intensity referral interventions. Our primary outcome is Veterans' connections to new resources to address unmet needs. Additional outcomes include unmet need reduction, adherence (medications, ambulatory care appointments), utilization (preventable hospitalizations, urgent care), and clinical outcomes (blood pressure, glycemic control).

# 3.0 Objectives

We will compare outcomes among Veterans with or at risk for CVD at three VA sites randomized (at the site-level) to one of three arms: 1) unmet needs screening only, 2) screening + provision of tailored resource sheets to address identified unmet needs, or 3) screening + tailored resource sheet + social worker support. We will quantitatively examine associations of unmet needs with baseline and follow up outcomes, assessing the impact of varying intensity referral approaches. We will also qualitatively examine stakeholder perspectives about the barriers and facilitators to identifying and addressing unmet needs to provide insight into the relative success of each study arm. Specific aims are:

**Aim 1**: Describe the prevalence and distribution of nine unmet needs (housing, food insecurity, utility insecurity, transportation, legal needs, employment, safety, social isolation, stress), and identify their associations with baseline sociodemographic characteristics, adherence, utilization and clinical outcomes.

Aim 2: Compare the effectiveness of varying intensity referral strategies to address unmet needs on the primary outcome of connection to new resources to address unmet needs, and on secondary outcomes of post-intervention change in unmet needs, adherence, utilization, and clinical outcomes. H1. Based on Maslow's model, we hypothesize that referrals (and more so for those enhanced by SW support) will increase the likelihood of patients connecting to new resources to address unmet needs (primary outcome), which may then have positive sequential effects, with reduced unmet needs, increased adherence, decreased urgent care/preventable utilization, and ultimately, improved clinical outcomes.

**Aim 3**: Identify barriers and facilitators to Veterans' connecting with resources to address unmet needs and getting needs met, and explore potential explanatory factors related to the relative success of each study arm.

This project addresses HSR&D priorities of health equity and population health, the Office of Social Work's goal to link Veterans with resources and services in support of treatment goals, the Office of Patient Centered Care and Cultural Transformation's priority to enhance the physical, emotional, and social well-being of the whole person, the Office of Health Equity's priority to address unmet needs to ensure health equity, and the Office of Primary Care's aim to provide personalized, comprehensive and coordinated care. Findings from this study will provide crucial information to inform future efforts to identify and address Veterans' unmet needs.

## 4.0 Resources and Personnel

#### PERSONNEL: VA BOSTON HEALTHCARE SYSTEM, BOSTON, MA

**Deborah Gurewich, Ph.D., Principal Investigator**, (8/8th VA). Dr. Gurewich is an Investigator at the Center for Healthcare Organization and Implementation Research (CHOIR) based at the Boston VA Healthcare System (HCS). Dr. Gurewich will have overall responsibility for leading and directing the study including coordinating all study personnel, leading weekly project meetings, and communicating with our operational partners. She will also oversee the research staff at each study site, which will include ensuring that staff are trained on the intervention and convening standing meetings with each site to track and monitor the trial implementation. She will have access to protected health information (PHI).

Amy Rosen, PhD co-Investigator (8/8th VA). Dr. Amy Rosen is a Senior VA HSR&D Research Career Scientist based at CHOIR Boston with over 30 years of experience as a health services researcher. Dr. Rosen has extensive experience in collaborating with multiple VA sites, conducting and analyzing survey data, using large VA administrative databases (including data from the Corporate Data Warehouse), and in conducting advanced hierarchical regression models and other multivariate analyses. She will advise Dr. Gurewich on the quantitative methods.

**Barbara Niles, PhD co-Investigator** (8/8th VA). Dr. Niles is a clinical psychologist in the Behavioral Science Division of the National Center for PTSD at VA Boston Healthcare System. She is an experienced clinical trialist with deep experience in the design and management of clinical trials, and in implementing such trials in VA clinical settings. Dr. Niles will advise Dr. Gurewich on the design, implementation and over-sight of the clinical trial.

Amy Linsky, MD, MSc co-Investigator/Local Site Investigator (8/8th VA). Dr. Linsky is an Investigator at Boston CHOIR and a board-certified internist in the section of General Internal Medicine at VA Boston Healthcare System. She has a dual role on the project. As co-I, she will provide clinical input on how SDoH affects the provision of care and health care utilization and outcomes, and advise on current practices within VA for identifying and addressing SDoH and interpreting study findings within this context. In her second role, se will serve as the Local Site Investigator for the Boston RCT site and in that capacity be responsible for ensuring recruitment and retention of study participants at VA Boston. She will have access to PHI.

Hannah Friedman, PhD., co-Investigator (8/8ths VA). Dr. Friedman is a post-doctoral fellow at Boston CHOIR. As part of her fellowship plan, she will assist the PI with data analysis in Aims 1, 2, and 3 and supporting dissemination efforts. She will have access to PHI.

Risette (Zoe) MacLaren, MSc, Project Manager (8/8ths VA). Ms. MacLaren is a senior project manager at Boston CHOIR. She will coordinate with project staff across the sites, maintain IRB approval and regulatory documents, ensure that database development and data analyses are on track, and oversee the maintenance of study data in a secure fashion. Ms. MacLaren will attend all project meetings and keep study records.

**Daniel J Sturgeon, MS, Data Analyst** (8/8ths VA). Mr. Sturgeon is a program analyst at Boston CHOIR. He will be responsible for identifying eligible participants in Y1. Working closely with Dr. Li, he will be responsible for developing the analytic data sets, which will involve pulling data from VA's Corporate Data Warehouse (CDW) and merging with primary data (the two rounds of unmet need screening data and the 8-week follow-up survey). He will also be responsible for all programming related to executing the analytic models. He will have access to PHI.

**Alexa Silva, MSW** (8/8ths VA). Ms. Silva is a master's level social worker (MSW) on the study team at the Boston VAMC for Year 2 only. She will be based at the Boston study site and responsible for providing SW support services to Veterans randomized to the third study condition. She will have access to PHI.

Rory Ostrow, MPH, Research Assistant (8/8ths VA). Mr. Ostrow is a Boston CHOIR Research Assistant. He will assist Ms. MacLaren in key aspects of the day-to-day management of the project, including the IRB and related DART applications, and subsequent amendments as needed. He will also assist with developing the resource sheets in Boston and oversee the resource sheet development in Charleston and Philadelphia. He will work closely with Dr. Gurewich in managing the qualitative data, as well as coding and analysis of the qualitative data. He may also conduct some of the qualitative interviews, as needed. He will have access to PHI.

Kathleen Codair, BS Research Assistant (8/8ths VA). Ms. Codair is a Research Assistant at VA Boston CHOIR. She will be based at the Boston clinical site and responsible for administering the unmet need screens, providing resource sheets to trial participants who identify unmet needs, and conducting the 8-week follow-up survey to determine if Veterans connected to services or not. She may also conduct qualitative interviews with select Veterans participating in the trial and representatives of VA programs and community organizations. She will only be involved in Boston site research activities. She will have access to PHI.

PERSONNEL: EDITH NOURSE ROGERS MEMORIAL VETERANS HOSPITAL, BEDFORD, MA

Barbara Bokhour, Ph.D., co-Investigator (8/8ths VA). Dr. Bokhour is an investigator and Director at Bedford CHOIR. Dr. Bokhour has led studies that identified the importance of Veterans' social context in managing their CVD, as well as developed a stories-based intervention whereby African-American Veterans who had successfully managed their hypertension described strategies to reduce their CVD risk. She will advise on all elements of the study.

Gemmae Fix, PhD, Local Site Investigator (8/8ths VA). Dr. Fix is an Investigator at Bedford CHOIR. She is supported by a Career Development Award through HSR&D CDA 14-156, with Drs. Bokhour as mentor. She is exploring the effects of SDoH in older Veterans with HIV and aging-related comorbidities like hypertension and CVD. She has expertise in qualitative methods. She will be a key member of the Aim 3 qualitative team, contributing to finalizing the interview guides and assisting with data coding and analysis. She will also be involved in all study planning, and review and interpretation of findings.

**Mingfei Li, Ph.D., co- Investigator** (IPA). Dr. Li is a Statistical Scientist at Bedford CHOIR and a Professor of Mathematics at Bentley University in Waltham, MA. Dr. Li has experience with multilevel modeling, multiple regression, and structural equation modeling, as well as mixed-methods approach. She will be responsible for the statistical modeling for this project. She will have access to PHI.

PERSONNEL: CORPORAL MJ CRESCENZ VA MEDICAL CENTER, PHILADELPHIA, PA

Melissa Dichter, PhD, MSW Local Site Investigator (8/8ths VA). Dr. Dichter is the Associate Director and Core Investigator at the U.S. Department of Veterans Affairs Center for Health Equity Research and Promotion (CHERP) in Philadelphia, PA, and an Assistant Professor at the University of Pennsylvania Perelman School of Medicine, Department of Family Medicine and Community Health. She has strong working relationships with members of the investigative team as well as operations

partners. She will be responsible for hiring and supervising local staff, and ensuring recruitment and retention of study participants at the Philadelphia VA. She will also be responsible for obtaining necessary regulatory approvals for the site, participating in team meetings, helping to interpret findings and prepare reports for dissemination. She will participate in calls with the rest of the leadership team and assist in analyses and dissemination of findings. She will have access to PHI.

Catherine Westerduin, MSW, Social Worker (8/8ths VA). Ms. Westerduin will serve as master's level social worker (MSW) at the Philadelphia VAMC for Year 2 only. She will be based at the Philadelphia study site and responsible for providing SW support services to Veterans randomized to the third study condition. Ms. Westerduin will have access to PHI.

Aneeza Agha, MA, Research Assistant (WOC, University of PA). Ms. Agha is based at the Philadelphia VAMC and will work with Ms. Morawej on administering the unmet need screens, providing resource sheets to trial participants who identify unmet needs, and conducting the 8-week follow-up survey to determine if Veterans connect to services or not. She may conduct qualitative interviews with select Veterans participating in the trial and representatives of VA programs and community organizations. She will assist with creating and maintaining resources sheets at this site. She will have access to PHI.

**Sabrina Morawej, MPH, Research Assistant** (8/8ths VA). Ms. Morawej is based at the Philadelphia VAMC and will work with Ms. Agha on administering the unmet need screens, providing resource sheets to trial participants who identify unmet needs, and conducting the 8-week follow-up survey to determine if Veterans connect to services or not. She may conduct qualitative interviews with select Veterans participating in the trial and representatives of VA programs and community organizations. She will assist with maintaining resource sheets at this site. She will have access to PHI.

## PERSONNEL: RALPH H JOHNSON MEDICAL CENTER, CHARLESTON, SC

Kelly Hunt, PhD, MSPH Local Site Investigator (8/8ths VA). Dr. Hunt is an investigator at Charleston VA Health Equity and Rural Outreach Innovation Center (HEROIC), a Center of Innovation (COIN) and a Professor in the department of Public Health Science at the Medical University of South Carolina. She will be responsible for hiring and supervising local staff and to ensure recruitment and retention of study participants from the Ralph H Johnson VAMC. She will also be responsible for obtaining necessary regulatory approvals for the site, participating in team meetings, helping to interpret findings and prepare reports for dissemination. She will participate in calls with the rest of the

leadership team and assist in analyses and dissemination of findings. She will have access to PHI.

**Tyler Singleton, MSW** (8/8ths VA). Ms. Singleton is a master's level social worker (MSW) at the Charleston VAMC for Year 2 only. She will be based at the Charleston study site and responsible for providing SW support services to Veterans randomized to the third study condition. She will have access to PHI.

Lauren Fanning, MPH, Research Assistant (8/8ths VA). Ms. Fanning will be based at the Charleston VAMC and will administer the unmet need screen, provide resource sheets to trial participants who identify unmet needs, and conduct the 8-week follow-up surveys to determine if Veterans connect to services or not. She may also conduct qualitative interviews with select Veterans participating in the trial and representatives of VA programs and community organizations. She will assist with maintaining resource sheets at this site. She will have access to PHI.

#### SERVICES PERFORMED BY CONTRACTORS

We will use Alpha Transcription to transcribe the qualitative interviews.

# 5.0 Study Procedures

# 5.1 Study Design

To assess the efficacy of systematic S&R, we propose a two-phase, three-year mixed methods study (Phase One: quantitative, Phase Two: qualitative) to systematically screen Veterans with or at risk for CVD for nine unmet needs, characterize the prevalence of unmet needs and association with outcomes, and compare the effects of two different referral interventions of varying intensity on multiple outcomes.

In **Phase One (Aim 1)** we will survey Veterans about their unmet needs (N=1760) and conduct quantitative analyses of survey, administrative, and clinical data to characterize the prevalence of unmet needs and their association with baseline outcomes (adherence, utilization, and clinical). In **Phase One (Aim 2)**, we will implement a three-armed RCT at three VA sites to compare outcomes among Veterans with one or more unmet needs (N=880) randomized within each site to one of three intervention arms. Trial participants will participate in three surveys, all administered by phone: 1) an initial index unmet need survey; 2) an eight week follow-up survey to assess if participants connected to any new resources since the index screen and if so, to which one(s); and 3) six months after the initial index screen, the unmet need survey will be administered again.

We have the following study arms: 1) Unmet needs screening and provision of a post card with a generic list of VA resources (hereafter: "Screening" arm), 2)

Screening and provision of a post card with a generic list of VA resources plus provision of a tailored Resource Sheet listing available resources to address identified unmet needs (hereafter: "Awareness" arm), or 3) Screening and provision of generic list of VA resources plus provision of a tailored Resource Sheet plus research team SW-supported referral to assist with connection to resources for unmet needs (hereafter: "Assistance" arm). Quantitative analyses will longitudinally compare the effects of the two referral approaches of varying intensity and a generic intervention on the primary outcome of connections to new resources and secondary outcomes of reduction in unmet needs, adherence, utilization, and health outcomes. See **Appendix A** for a more detailed description of the intervention and approach to randomization.

In **Phase Two (Aim 3)**, we will conduct qualitative interviews with a purposeful sample of Veterans (N=60) and representatives of the VA- and community-based programs to which Veterans are referred (N=15). The interviews are designed to understand the conditions that facilitate and impede Veterans' connection to resources and unmet need reduction, and to identify potential explanatory factors related to the relative success of the interventions. We will follow standard qualitative methods for data collection, coding, and analysis.

# Risk to Subjects

We are implementing a non-invasive behavioral intervention by screening and referring Veterans in some study arms to resources to address unmet needs, and in one arm, connecting Veterans with a social worker to support them in connecting to resources. Potential risks are minimal and would primarily involve loss of confidentiality, as follows.

#### **Phase One**

- Quantitative Data (Administrative Databases): Given that we are using
  existing data sources, there will be no direct health risks to subjects as a
  result of the proposed research. The risks associated with the use of these
  existing data sources would be due to possible breaches of privacy and
  confidentiality.
- Quantitative Data (Surveys): Potential risks may include breaches of privacy and confidentiality. Veterans answering the survey items may also feel inconvenienced and/or uncomfortable answering questions about unmet needs and connection to resources to address unmet needs. Finally, Veterans randomized to the least referral-intense arm (screening-only) could get frustrated with this assignment if they want more assistance with identified needs than this arm offers.


#### Phase Two

 Qualitative Data (Interviews): For the interviews with Veterans and representatives of organizations providing resources to help Veterans address unmet needs, potential risks may include breaches of privacy and confidentiality, inconvenience, as well as discomfort (in the case of Veterans) answering questions about unmet needs and accessing resources.

## **Adequacy of Protection from Risk**

We have conducted a wide array of studies that require us to make careful use of confidential information. In addition, the VA Boston HCS and CHOIR have systems, oversight, experienced personnel, and organizational cultures that support the appropriate use of confidential information, thus helping to further minimize and protect study subject from potential risks. Collected data will be used only for research purposes and identifiers will be removed from all data files, which will only be identified with a study identifier (except for audio recordings which include voice as an identifier). Reported results will not contain any individual identifiers. Research records will be destroyed in accordance with the VHA Records Control Schedule (RCS). Paper files will be shredded. Research data maintained on electronic storage and memory devices such as computers, laptops, and CDs will be destroyed in a way it cannot be retrieved.

#### **Phase One**

Quantitative Data (Administrative Databases): Only the Principal Investigator and study team members conducting data analyses will have access to the secondary data obtained from the national VA databases. We will store and analyze secondary data on two servers located at: 1) the VA Informatics and Computing Infrastructure (VINCI) and 2) VA Boston HCS. The secondary data obtained through the CDW will be stored and analyzed on VINCI, a VA proprietary data storage space that allows data analysis to occur in a virtual environment. This has the benefit of allowing data analysis to occur from VAencrypted desktops and laptops. The VINCI Workspace is a VA-secure, virtual computing environment. It is accessed through a single secure gateway for all users. The virtual environment is maintained from a central management server and provides a separate path for secure file transfer for controlling the security of the Workspace to prevent the removal of data. We will request permission for the data analyst to export datasets associated with this study to the VINCI server. Data will be uploaded to VINCI which allows both data storage space and data analysis to occur in a virtual secure environment providing even more protection from breach of confidentiality.

Secondary data may also be stored and analyzed on the VA Boston HCS server behind the firewall. Access to the computer systems is restricted and password protected. All research computers are located in locked offices and computers are password protected. Access to CHOIR offices is restricted. All space accessible to the public is separated from research offices.

For all secondary data, we will take all necessary steps to protect privacy and confidentiality, in accordance with VA regulations and other applicable laws. All information on individuals will be kept confidential. Consistent with HIPAA regulations, we will use scrambled identifiers (when available) to allow linkages across files while protecting an individual's identity or we will de-identify the datasets. Only project personnel will have access to the data.

Quantitative Data (Surveys): We will construct a secure, password protected database in VA REDCap (to which we already have access as a team) to input the survey data. Survey data will be stored in this secure database at VA Boston and all personnel who need access will be able to connect to the server. Data will be cleaned and checked for accuracy by the project manager and data analyst. Mishandling of research data would compromise participant confidentiality. Thus, all possible measures will be taken to assure Veteran confidentiality. In addition, we will construct a secure, password protected database to create a record of study participants and those who have opted out of the study, using scrambled SSNs. This will be stored on a secure VA Boston server.

To protect against risks associated with a Veteran getting upset during any of the survey processes, the RA will be trained to deal with difficult situations and remind participants that they may decline to answer any question or discontinue the survey at any time. Additionally, the research SW at each site will be on-call to assist as needed. In the rare instance that during the intervention either the RA or SW encounter unknown risks affecting participants health and welfare, they will advise the participant to contact their primary care team and with participant approval also notify the care team directly. If a participant indicates that he or she is having suicidal or homicidal thoughts, the RA and SW will be trained to offer the Veterans Crisis Line and a warm hand-off using established protocols (see **Appendix B** for warm hand-off protocol), and with participant approval also notify the care team directly.

To protect against risks associated with Veterans who are unhappy about the condition to which they are randomized, we will take several steps to minimize this risk: 1) As part of the informed consent process, we will be explicit about the three study arms, that we cannot predict which arm a Veteran will be randomized

to; and 2) we will be clear that this a research study, which means that information we gather from Veterans will not be shared with their care team but that participants are welcome to follow-up with their care team at any time during their participation in the study. The RA will also be prepared to provide the care team phone number to the Veteran, if needed.

#### Phase Two

Oualitative Data (Interviews): To protect against risks related to privacy and confidentiality, we will use VA computers to take notes and a VA Boston HCS IRB and Information Security Officer approved audio recorder and software (SpeechExec Pro Dictation and Transcription Software) when conducting the telephone interviews. Interviews will be digitally audio-recorded, with the permission of each Veteran. If a subject asks us to not record a portion of the interview, the recorder will be turned off immediately. The list of individuals who participate in interviews will be kept on the VA Boston server and will be recorded in a document that is password protected with restricted access to the members of the study team working on the qualitative data collection and analysis. Notes that are taken will be de-identified. Encrypted recordings will be emailed to the study team. The study team will store recordings on a secure VA server and will be password protected. All names and places mentioned will be deleted to protect confidentiality. De-identified audio-recordings will be transcribed by Veterans Command Transcription, a premier service provider for the VA. Transcribed interviews will be imported into a qualitative software program designed for maintaining and analyzing qualitative data.

To protect against inconveniencing participants, we will restrict the length of the interviews to 45-60 minutes. To protect against risks associated with a Veteran getting upset during the interview, the RA will be trained to deal with difficult situations and remind participants that they may decline to answer any question or discontinue the interview at any time.

#### **Potential Benefits**

- Veterans will receive a post card that includes a list of VA crisis and homeless hotlines that can be immediately useful.
- Veterans will receive information about specific VA and community programs that can also be immediately useful.
- We will develop a screening tool to identify unmet needs and identify which approach to referral is better and under what conditions at helping Veterans connect to resources and at affecting outcomes. Our tools and

the findings can be used in the field to implement screening and referral processes to address unmet needs, and by other researchers studying this issue.

- Our study will identify the full burden of unmet needs among Veterans as well as which needs and clusters of needs are most impactful with respect to outcomes, information that can inform how and where VA targets resources to address unmet needs.
- If our study finds that systematic screening and referral for unmet needs is associated with improved outcomes, our study will establish the needed evidence base for more wide-spread adoption of this practice, which has the chance to benefit all VA-enrolled Veterans who experience unmet social needs.

## Safety and Data Monitoring Plan

Per FOA/RFA instructions, given that we are proposing a multisite intervention trial with human participants, HSR&D DSMB oversight is required. DSMB approval is accomplished by an independent review board chartered by HSR&D that meets at specified intervals and requires routine reporting from the PI. The PI will follow a specific Data and Safety Monitoring Plan and per HSR&D program guidelines, has submitted a Data Analysis Plan (DAP) as part of the Just-In-Time (JIT) compliance process. Studies are generally not allowed to begin until DSMB approval of the DAP has been provided. Currently, the DSMB meets on annual basis (generally in the early spring) but can request (or review) studies more frequently (if they determine that to be appropriate). The PI will receive a letter regarding the DSMB's determination after the meeting, including any concerns and follow-up actions; the PI will then submit these letters to VA CIRB.

We anticipate minimal risk, as the proposed intervention is survey-based and providing resources but once the study is underway, study staff and investigators will monitor any adverse events and immediately report any adverse events to the DSMB. The Principal Investigator (PI) and project manager (PM) will routinely audit the data for accuracy and make any necessary corrections to ensure data reliability and accuracy. In addition, the PI and PM will review the plans for and implementation of subject recruitment and enrollment, to ensure adequate recruitment progress and that recruitment milestones are met. Recruitment problems will be identified and addressed and if necessary, sites without adequate enrollment will be replaced.


Site monitoring progress reports will be submitted to the DSMB and other regulatory bodies (e.g., CIRB) as requested and/or required. As described in Section 5.1.b (Protection Against Risk), we will monitor every step of our recruitment procedures, survey data collection, and interviews to ensure that the confidentiality and privacy of our study populations are protected. Should we receive any negative feedback from research subjects or have any unexpected serious or adverse events, we will report this information to the DSMB, VA Central IRB, and local R&D offices immediately.

In the unlikely event of a breach of confidentiality, the incident will be documented and reported to the DSMB, VA Central IRB and R&D immediately, as will any incident of protocol deviation. We will ensure the rights to privacy, confidentiality and safety are maintained.

There is no safety condition that would trigger immediate suspension of the study.

# **Study Population**

Phase One (Aim 1): The study population will be comprised of Veterans from the primary care (PC) clinics of three VA medical centers: 1) VA Boston Healthcare System; 2) Corporal Michael J. Crescenz VA Medical Center (Philadelphia); and 3) Ralph H. Johnson VA Medical Center (Charleston). Veterans with, or at risk for, cardiovascular disease (CVD) who had at least 1 PC visit in the prior year, will be eligible for the study, to ensure that included Veterans are at least minimally engaged in VA care. We define CVD patients as those with International Classification of Disease 10 (ICD10) diagnoses indicating coronary artery disease, cerebrovascular disease, or peripheral artery disease, and patients with CVD risk factors as having diagnoses of hypertension, diabetes mellitus (DM), or hyperlipidemia. We will exclude Veterans who have 1) impaired decision-making, and/or 2) are illiterate or have limited or no English proficiency.

**Phase One (Aim 2):** The study population will be comprised of the subset of subjects in Aim One who report having one or more unmet needs.

**Phase Two (Aim 3):** The study population includes a purposeful sample of two stakeholder groups: 1) Veterans who participate in trial, and 2) representatives of the VA programs and community resources that Veterans are referred to as a result of the intervention.

Veterans: We will seek three Veteran types: Veterans who did not connect
to new resources; Veterans who connected to new resources but did not
have their unmet needs met, and Veterans who connected to new
resources and had their needs met. This sampling plan will allow us to
understand the conditions that facilitate or impede a Veteran connecting to

resources, as well as the conditions under which resources do or do not address a Veteran's needs. We will not exclude any subjects based on gender, race, or other classes (e.g., disabilities).

VA and Community Program Representatives: We will seek up to five of
the most frequently used programs at each study site (15 total). By
concentrating on the most highly used programs, this sampling plan will
allow us to understand the experience of programs more likely to "feel" the
effects of the intervention.

#### 5.2 Recruitment Methods

Step 1 (determine potential eligibility based on existing administrative data): The study will begin with a 12-month retrospective baseline period in which Veteran clinical eligibility (i.e., diagnosis of CVD or CVD-risk) will be determined using data from CDW. We will not exclude any Veterans based on race, gender, or other classes (e.g., handicapped). We will exclude two classes of Veterans: 1) those with impaired decision-making and 2) those who are illiterate or have limited or no English proficiency. This initial step involves secondary data analysis only; we will not recruit Veterans as subjects for use of secondary data; we will request a HIPAA Waiver of Authorization for this step.

Step 2 (initial outreach by mail to potentially eligible participants): For the next 12 months and on a weekly basis, the study Data Analyst will produce a primary care appointment list of eligible Veterans at each study site using data from CDW. In advance of an eligible Veteran's appointment, the research team will mail the Veteran the following documents:

- A Cover Letter briefly describing the study and inviting participation (see Appendix C);
- A Study Fact Sheet detailing the elements of informed consent and describing the study in more detail including that participants will complete a brief survey and based on the survey results, those deemed eligible for the RCT will be randomized to one of three study arms, while those deemed not eligible, will be done with the study after completing the initial survey (see Appendix D);
- A post card that includes phone numbers for the Veteran's VA Medical Center, VA Veterans Crisis Line, and National Call Center for Homeless Veterans (see Appendix E);
- An opt-out postcard (postage included) that will explain that the Veteran is
  eligible for the initial phase of the study and may be eligible for the
  subsequent phase, an RCT; indicate that if they are interested in

potentially participating that an RA will contact them by phone in advance of the Veterans upcoming PCP appointment, and; if they are not interested to return the opt-out card within 3 days of receiving it (see **Appendix F**).

Step 3 (phone follow-up to recruit, consent, and screen for eligibility): The research team will provide the final list of site-specific eligible Veterans who did not return an opt-out card to the RA situated at each study site. Guided by a phone script (see **Appendix G**), the RA will contact these Veterans by phone up to three weeks following the opt-out card mailing (making up to 5 attempts if they cannot reach the Veteran) to: 1) describe the study, 2) request participation, including potential randomization to one of three study arms if deemed eligible following the initial index screen, participation in subsequent surveys, and possible contact by phone to invite participation in a qualitative interview; and 3) obtain verbal consent. The RA will review the elements of informed consent and answer any questions the potential respondent might have. Among Veterans who verbally consent to participate, the RA will administer the index unmet need screen and, if Veteran is eligible for the RCT (i.e., 1 or more unmet needs) randomize them to one of the three trial arms using the sealed opaque envelope program (see **Appendix A** for details).

Step 4 (recruitment for qualitative interviews; Veterans): Among study participants, we will purposefully sample 60 Veterans to participate in qualitative interviews. Sample selection and recruitment will be conducted on a rolling basis after the 6-month unmet needs re-screen is completed. The study RA will phone selected Veterans, ask for participation in an interview, and among those who accept, schedule an interview time. Note: As part of the RCT informed consent process, participants will be told that they may be contacted by phone to participate in a qualitative interview, which we believe eliminates the need to mail opt-out cards prior to contacting Veterans by phone for this phase of the study. During this initial call we will not re-consent participants but will review and remind potential participants of the purpose of the interviews and the elements of informed consent.

Step 5 (recruitment for qualitative interviews; Agency representatives): We will also seek a purposeful sample of representatives of the VA and community programs that Veterans are referred to as a result of the intervention. Potential interviewees will first be contacted by email or phone (dependent on contact information available in VA Outlook and community agency websites) to assess their interest in being interviewed for the project. Each potential interviewee will be emailed a letter of invitation from the site PI (see **Appendix H** for Resource Representative Recruitment Email). The letter will contain all the elements of

consent: the risks and benefits of the study, confidentiality procedures, study personnel to contact regarding questions and concerns (including contact numbers for the VA Central Institutional Review Board), that participation is voluntary, and that participating or not participating in the interview will not affect their VA appointment (in the case of VA program representatives) or their organizational relationship with the VA (in the case of community program representatives). If a potential interviewee expresses interest in participating, we will use both email and phone to schedule an interview with the participant. A member of the study team will then review the letter before conducting an interview with any potential interviewee. Participation in the interview will be an indication of consent.

## 5.3 Informed Consent Procedures

Phase One (Aims 1 and 2): We will not recruit Veterans as subjects for use of secondary data given the minimal risks associated with the study. We will adhere to IRB requirements for informed consent and request a HIPAA waiver of authorization.

Phase One and Two (Aims 1, 2, and 3): The elements of informed consent will be provided in writing and orally, but we will seek a waiver of documentation of informed consent because the recruitment and informed consent process will be conducted entirely by phone, and we believe study poses no more than minimal risk.

To ensure consistent and thorough administration of the informed consent process for this study, the local RAs and investigators will be trained by the PI on the informed consent process and will conduct mock informed consent sessions with the PI prior to performing the informed consent process with patients. Site investigators and RAs will also be trained on the importance of allowing sufficient time for participants to consider the information provided and providing time and opportunity for the participants to ask questions and have those questions answered in order to inform their decision about whether to participate or not. We will conduct periodic internal audits of the informed consent process to ensure informed consent protocols are followed. These audits will take place weekly at the start of the outset of the study (i.e., first month of the trial) and then reduce in frequency as the study continues but will be at least two additional times over the remaining 11 months of the trial.

#### 5.4 Inclusion/Exclusion Criteria

Our study population will be comprised of Veterans from the primary care (PC) clinics of three VA medical centers: 1) VA Boston Healthcare System; 2)

Corporal Michael J. Crescenz VA Medical Center (Philadelphia); and 3) Ralph H. Johnson VA Medical Center (Charleston). Note: There is a 4<sup>th</sup> site involved in this study (Bedford) but we are not identifying and recruiting Veterans from this site. Veterans with, or at risk for, cardiovascular disease (CVD) who had at least 1 PC visit in the prior year, will be eligible for the study, to ensure that included Veterans are at least minimally engaged in VA care. We define CVD patients as those with International Classification of Disease 10 (ICD10) diagnoses indicating coronary artery disease, cerebrovascular disease, or peripheral artery disease, and patients with CVD risk factors as having diagnoses of hypertension, diabetes mellitus (DM), or hyperlipidemia. We will not exclude any patients based on gender, race, or other classes (e.g., disabilities). We will exclude patients with impaired decision-making capacity and who are illiterate or have limited or no English proficiency.

Among study participants, we will also recruit a purposeful sample of Veterans who participated in the trial as well as representatives of the VA and community programs to which participants are referred as a result of the trial. For the Veteran interviews, we will seek three Veteran types: Veterans who did not connect to new resources; Veterans who connected to new resources but did not have their unmet needs met, and Veterans who connected to new resources and had their needs met. For the VA and community program representatives, we will seek up to five of the most frequently used programs at each study site. We will not exclude any potential respondents for the qualitative interviews based on gender, race, or other classes (e.g., handicapped).

# **5.5 Study Evaluations**

RCT participants will be asked to complete three brief surveys over a 6-month period. A small sub-set of participants will additionally be invited to participate in qualitative interviews.

Index Unmet Need Screen (survey #1): We will assess unmet needs among trial participants based on the index screen (administered prior to randomization). See **Appendix I** for the Index Unmet Need Survey.

<u>Eight-Week Follow-Up Survey (survey #2):</u> Eight weeks after the index screen, the RA will conduct phone follow-up with each Veteran to assess if they connected to any new resources in the intervening time and if so, to which one(s). See **Appendix J** for the Eight-Week Follow-Up Survey and accompanying phone script.

<u>6-Month Unmet Need Re-Screen (survey #3</u>): Six months after the index screen and by phone, the RA will re-administer the unmet need survey modified slightly

to exclude questions related to preferences for assistance (see **Appendix K** for the Six-Month Unmet Need Survey and accompanying phone script). We will define unmet need reduction in two ways: 1) one or more of baseline unmet needs no longer identified as an unmet need at the 6-month re-screen; and 2) percentage of baseline needs not reported as unmet needs at 6-month rescreen.

Qualitative Interviews with Veterans: Among study participants, we will purposefully select and recruit 60 Veterans to participate in qualitative interviews. The interviews are designed to understand the conditions that facilitate or impede a Veteran connecting to resources, as well as the conditions under which resources do or do not address a Veteran's needs. The RA at each study site will conduct the interviews. See **Appendix L and M** for the Veteran Interview Guides and accompanying phone scripts).

Qualitative Interviews with Representatives of VA and Community Resources: To understand how VA- and community-based programs experience the intervention, we will interview a purposeful sample of the VA- and community-based programs that trial participants used as a result of the intervention. The RA at each study site will conduct the interviews. See **Appendix N** for the Resource Representative Interview Guide and accompanying phone script.

## 5.6 Data Analysis

## **Study Sample and Power Analysis**

We aim for a total of 880 Veterans enrolled in the RCT (293/arm) based on power analyses provided below. Based on the study team's prior primary care-based studies with a similar recruitment approach, we anticipate 80% of patients approached to complete the index screen will participate. Based on pilot data from the Bedford MA VA where 78% of Veterans reported one or more needs, we then conservatively estimate that 50% of Veterans screened will report at least one of the nine unmet needs for which we will screen.

Thus, to yield a final sample of 880 Veterans with at least one unmet need enrolled in the study, we anticipate needing to approach 2200 eligible Veterans (733/site, or ~3 patients/day/site) i.e., of 2200, 80% (1760) will agree to participate in the study and of these, 50% (880) will have one or more unmet needs and be eligible for the RCT. If the participation rate or proportion of Veterans reporting at least one unmet need is lower than expected, we will increase the number of Veterans that we approach. We reviewed VA administrative data to determine the anticipated weekly count of Veterans eligible per site to participate in the study and there are more

26

than enough eligible Veterans to approach for additional screening if needed. We also anticipate drop-out rates at the 8-week follow-up survey to assess connection to resources and the 6-month unmet needs rescreen, respectively. Though the study team's prior study achieved a 65% follow up participation rate, here we conservatively anticipate a 50% participation rate for both the 8-week follow-up survey and the 6-month rescreen, reducing the sample for the three arms first to 440 Veterans total and then to 220 Veterans total.

Statistical Power for Aim 1: With a sample of N=1760 Veterans completing the index unmet needs screening, we will have 80% power to detect small effect sizes (f2=.01; OR=1.47) using 2-tailed significance tests at the  $\alpha$ =.001 level if the intraclass correlation coefficient (ICC) (for the nesting of patients within sites) is negligible, or medium effect sizes (f2=.15; OR=4.07) even if the ICC is as high as .02 for testing associations between the presence of each unmet need and sociodemographic, adherence, utilization, and clinical (BP only) variables. HbA1c is anticipated to be a relevant clinical outcome for only 40% of the sample; for HbA1c, we will have 80% power to detect small effect sizes (f2=.03; OR=1.84) using 2-tailed significance tests at the  $\alpha$ =.001 level if the ICC is negligible.

Statistical Power for Aim 2: The power analysis for Aim 2 focused on the primary outcome of connection to resources to address unmet needs. The sample size was determined based on previous research outside VA which found that individuals who completed a screening and referral intervention were 15% more likely (adjusted Odds Ratio (aOR)=2.1) to have enrolled in a new community resource to address unmet needs postreferral compared to patients in the non-intervention arm. In the present study, we will have 80% power to detect an effect of this size (aOR=2.1) across the three arms using 2-tailed significance tests at the  $\alpha$ =.05 level. even if we assume an attrition rate as high as 50% for the follow-up phone call at 8-weeks post-screen (retained N=440 across all sites and arms) and a conservative ICC value for patients nested within sites of .01. Previous empirical work found ICC values < .0001 when adjusting for a small number of covariates (e.g., race, marital status) to examine new connections to resources to address unmet needs; we intend to collect and use these covariates in the present study as well. Assuming an ICC value of .0001, we will have 80% power to detect an effect as small as an aOR=1.7 if we assume a 50% attrition rate for the 8-week follow-up phone call, or as small as an aOR=2.0 if we assume a 70% attrition rate. We based our attrition rate upon the study team's prior study where Veterans


had low incomes, high unemployment and low educational status, yet only 35% were lost to a follow-up interview.

## **Quantitative Data Analysis**

All data analysis will be conducted by study team members based in Boston. Dan Sturgeon is the study Data Analyst who will be responsible for developing the analytic data sets and all programming related to descriptive statistics and multivariate models. He will work closely with Mingfei Li, the statistician who will be responsible for developing the statistical models and overseeing the overall analytic approach. All analysis will be conducted on VINCI.

Aim 1: Describe the prevalence and distribution of nine unmet needs (housing, food insecurity, utility insecurity, transportation, legal needs, employment, safety, social isolation, stress), and identify their associations with baseline sociodemographic characteristics, adherence, utilization and clinical outcomes.

Our primary analysis for Aim 1 will be descriptive. We will use data obtained during the index screening (N=1760) to generate descriptive statistics (e.g., proportions, 95% confidence intervals (CIs) to characterize the prevalence and distribution of each of the nine unmet needs at baseline across all study sites. We will next conduct inferential analyses to examine associations between unmet needs and sociodemographic characteristics as well as baseline outcomes (i.e., adherence, utilization, and clinical outcomes drawn from CDW data in the 12-months before the index screening for each Veteran). Hierarchical Linear Modeling will be used to control for the nesting of patients within sites, and patient-level variables will be treated as random effects. Hierarchical Generalized Linear Modeling (HGLM) will be used as appropriate to handle binary variables. Variables found to have statistically significant associations with unmet needs will be entered into multivariable models to better understand the correlates of each need. Bonferroni-corrected significance levels will control for multiple comparisons.

Aim 2: Compare the effectiveness of varying intensity referral strategies to address unmet needs on the primary outcome of connection to new resources to address unmet needs, and on secondary outcomes of post-intervention change in unmet needs, adherence, utilization, and clinical outcomes

Our primary Aim 2 analysis will compare *connection to new resources* at 8-weeks post-index screen (our primary outcome of interest) across the study arms. HGLM will be used to control for the nesting of patients within sites. In all models, patient-level intercepts and slopes will be treated as random effects. We predict significantly greater connection to new resources in the ASSISTANCE arm

compared to the SCREENING arm, with the AWARENESS arm falling intermediate to these other two study arms.

Adherence, Utilization, and Clinical Outcomes. We will also conduct a series of secondary analyses to examine whether the study arms influence more distal outcomes, including adherence, utilization, and clinical outcomes. Specifically, to assess the impact of our intervention on more distal healthcare outcomes, we will use a difference-in-difference approach to examine whether changes from baseline at 6-months and 12-months post-referral differ across the three arms of our RCT (N=880). A series of HLM/HGLM analyses with patients nested within sites will examine differences in change from baseline across arms for the adherence, utilization, and clinical outcomes. As with the other analyses, all models will treat patient-level intercepts and predictors as random effects. We will have 80% power to detect small-to-medium effects (f2=.05; OR=2.28) across the three arms using 2-tailed significance tests at the  $\alpha$ =.05 level, even if we assume a conservative ICC value for patients nested within sites of .01. HbA1c is anticipated to be a relevant clinical outcome for only 40% of the sample and we anticipate missing HbA1c test data for 17% of these Veterans in the year following their index screen; thus, for HbA1c, we will have 80% power to detect small-to-medium effects (f2=.08; OR=2.71) across the three arms using 2-tailed significance tests at the  $\alpha$ =.05 level, even if we assume a conservative ICC value for patients nested within sites of .01.

Unmet Need Reduction: Similar analyses will be used to examine differences across our three study arms in change from baseline in the proportion of unmet needs among the sub-sample of participants who complete the re-screening at 6-months post-referral. Among this sub-sample (N=220, assuming attrition rates of 50% at both the 8-week and 6-month follow-up phone surveys), we will have 80% power to detect a small-to-medium effect (f2=.09; OR=2.94) across the three arms in terms of unmet need reduction using 2-tailed significance tests at the  $\alpha$ =.05 level, even if we assume a conservative ICC value for patients nested within sites of .01.

Differences in Intervention Effectiveness. In addition to examining how the S&R influences connection to new resources, we will conduct additional analyses to examine whether there is differential impact between the two referral arms (Awareness and Assistance) on connection to new unmet needs resources; unmet need reduction; and adherence, utilization and clinical outcomes among Veterans with certain unmet needs or with fewer unmet needs. While we predict that providing SW support (Assistance arm) will generally have a larger impact on outcomes than providing a Resource Sheet alone (Awareness arm), it would be beneficial to know if the Resource Sheet alone (or even the screening and

provision of generic list of resources) is sufficient to produce comparable changes in outcomes among Veterans with certain unmet needs or among Veterans with fewer unmet needs. If true, future implementation research could create tailored interventions that funnel the resources for more time- and cost-intensive referral strategies to only those Veterans who need it most.

Testing Conceptual Path. To the extent that we discover differences across intervention arms in any of our more distal outcomes, we will conduct exploratory analyses to test appropriate causal mediational paths as proposed in our conceptual model using a series of HLM/HGLM analyses (with patients nested within sites). That is, we will examine whether the impact of our intervention on more distal outcomes (e.g., BP) can be explained completely (or in part) by its impact on more proximal outcomes (e.g., connection to new resources, reduction in unmet needs). For example, if we find differences across study arms in reduction in unmet needs, we will test whether the effect of the intervention arm on reduction to new resources.

Examining marginal intervention effects over and above S&R occurring as part of usual care. Finally, given that Veterans may already be accessing resources for some unmet needs as part of usual care and related to existing screening for homelessness and food insecurity, we will conduct supplemental analyses to examine whether our intervention effects hold when controlling for use of VA SW services not attributable to the present intervention (e.g., services already being accessed separate from the study intervention). Although we will specifically be assessing connection to new resources following the S&R mechanisms in our three study arms, it is possible that individuals already connected to certain resources will be more likely to seek out additional support/resources (e.g., because they already have successful experiences using VA resources to meet certain unmet needs) or less likely to seek out additional support/resources (e.g., because they feel they already have the support they most need). Because VA screens for housing and food insecurity, Veterans may already be accessing resources for these. To examine whether the intervention has a significant impact on connection to new resources, unmet need reduction, and more distal health outcomes when controlling for use of VA SW services not attributable to the present study, we will conduct supplemental analyses that control for connection to resources associated with each of our nine unmet needs prior to enrollment in our intervention. Use of SW resources not attributable to our study will be measured via CPRS encounter forms, where SWs record encounters with patients, and from referral/consult documentation available in CPRS during the 12 months prior to the start of our intervention.


## **Qualitative Data Analysis**

Aim 3: Identify barriers and facilitators to Veterans' connecting with resources to address unmet needs and getting needs met, and explore potential explanatory factors related to the relative success of each study arm.

Transcripts will be initially coded using a priori constructs consistent with our conceptual model (Anderson Behavioral Health Model). A directed content analysis approach, allowing for new themes to emerge will be used. 17 As coding proceeds, new emergent themes will iteratively be identified, elaborated upon. and expanded based on team discussion. 18 New coding definitions may also be refined, and existing categories split and combined in the development of the coding matrix. This iterative process will eventually evolve to a point where all the existing categories will be sufficient to cover all new interview material that is obtained. The qualitative data analysis will be conducted by 3 study team members (Gurewich, Fix, Ostrow) and inter-rater reliability will be established using the "check-coding" process. 19 All coders will independently code the same interview transcripts, and initial reliability estimates between all pairs of coders will be computed. Coders will then meet to compare their coding, discuss areas of difficulty, and attempt to reach agreement. A new interview will then be independently coded by all, and the process will be repeated until a reliable level of agreement (>80%) is achieved across all coders. <sup>19</sup> After coding is complete, code output will be analyzed to identify themes within and across sample strata. All coding and analyses will be conducted using NVIVO qualitative analysis software.

# 5.7 Withdrawal of Subjects

There are not any anticipated circumstances under which subjects will be withdrawn from the research without their consent. Veteran participants may withdraw from the study at any time by telephone or email, which will be documented in the study files by the PI. Veteran participants can also stop any of the surveys – and for the relevant sub-sample, the interviews – at any time while they are happening.

# 6.0 Reporting

Dr. Gurewich will lead regular study team meetings and will formally query the study team specifically for any serious adverse events, unanticipated occurrences related to subject safety, breaches of study protocol or confidentiality. Study team members will also be directed to bring any such problems to the attention of the PI as they occur. The PI will report relevant

occurrences both to the Central IRB and the site R&D Committee per VA procedures.

# 7.0 Privacy and Confidentiality

The study will not disclose protected heath information. All information on individual subjects will be kept confidential on restricted server files behind the VA firewall. Collected data will be used only for research purposes and identifiers will be removed from all data files, which will only be identified with a study identifier (except for audio recordings which include voice as an identifier). Only study team members will have access to the secure file containing study data on encrypted VA served, and access will be removed for personnel when they are no longer part of the study through IT request. Study staff will be well trained to protect the privacy of study participants and prevent breaches of confidentiality. All study team personnel with access to sensitive patient data will stay current on required VA information security and privacy policy trainings. Reported results will not contain any individual identifiers. Research records will be destroyed in accordance with the VHA Records Control Schedule (RCS). Paper files will be shredded. Research data maintained on electronic storage and memory devices such as computers, laptops, and CDs will be destroyed in a way they cannot be retrieved.

#### 8.0 Communication Plan

All site approvals will be obtained in compliance with Central IRB procedures. For each site participating in the study, we will notify the Director prior to conducting research at his/her facility. Also, we will process any changes in the protocol, informed consent, or cessation of engagement in research for any sites in concordance with Central IRB procedures.

The PI will meet regularly with the study team, with local site co-Investigators participating via VANTS conference lines and Skype videoconferencing systems.

#### 9.0 References

Bibliography of cited literature

- 1. Frieden TR. A framework for public health action: the health impact pyramid. *Am J Public Health*. Apr 2010;100(4):590-5. doi:10.2105/ajph.2009.185652
- 2. McGinnis JM, Williams-Russo P, Knickman JR. The case for more active policy attention to health promotion. *Health Aff (Millwood)*. Mar-Apr 2002;21(2):78-93. doi:10.1377/hlthaff.21.2.78

- 3. Maslow AH. A theory of human motivation. *Psychological Review* 1943;50(4):370-96.
- 4. Kuh D, Hardy R, Langenberg C, Richards M, Wadsworth ME. Mortality in adults aged 26-54 years related to socioeconomic conditions in childhood and adulthood: post war birth cohort study. *BMJ*. 11/9/2002 PMC131184 2002;325(7372):1076-1080. Not in File.
- 5. Lawlor DA, Ronalds G, Macintyre S, Clark H, Leon DA. Family socioeconomic position at birth and future cardiovascular disease risk: findings from the Aberdeen Children of the 1950s cohort study. *AmJPublic Health*. 7/2006 2006;96(7):1271-1277. Not in File. doi:AJPH.2005.066290 [pii];10.2105/AJPH.2005.066290 [doi]
- 6. Lawlor DA, Smith GD, Ebrahim S. Association between childhood socioeconomic status and coronary heart disease risk among postmenopausal women: findings from the British Women's Heart and Health Study. *AmJPublic Health*. 8/2004 2004;94(8):1386-1392. Not in File. doi:94/8/1386 [pii]
- 7. Thurman WA, Harrison T. Social Context and Value-Based Care: A Capabilities Approach for Addressing Health Disparities. *Policy, politics & nursing practice*. Feb 2017;18(1):26-35. doi:10.1177/1527154417698145
- 8. Daniel H, Bornstein SS, Kane GC. Addressing Social Determinants to Improve Patient Care and Promote Health Equity: An American College of Physicians Position Paper. *Ann Intern Med.* Apr 17 2018;168(8):577-578. doi:10.7326/m17-2441
- 9. Havranek EP, Mujahid MS, Barr DA, et al. Social Determinants of Risk and Outcomes for Cardiovascular Disease: A Scientific Statement From the American Heart Association. *Circulation*. Sep 1 2015;132(9):873-98. doi:10.1161/cir.000000000000228
- 10. Garg A, Toy S, Tripodis Y, Silverstein M, Freeman E. Addressing social determinants of health at well child care visits: a cluster RCT. *Pediatrics*. Feb 2015;135(2):e296-304. doi:10.1542/peds.2014-2888
- 11. Gordon JA, Emond JA, Camargo CA, Jr. The State Children's Health Insurance Program: a multicenter trial of outreach through the emergency department. *Am J Public Health*. Feb 2005;95(2):250-3. doi:10.2105/ajph.2003.037242
- 12. Berkowitz SA, Hulberg A, Standish S, Reznor G, Atlas SJ. Addressing unmet basic resource needs as part of chronic cardiometabolic disease management. *JAMA internal medicine*. 2017;177(2):244-252. doi:10.1001/jamainternmed.2016.7691
- 13. Garg A, Marino M, Vikani AR, Solomon BS. Addressing families' unmet social needs within pediatric primary care: the health leads model. *Clinical pediatrics*. Dec 2012;51(12):1191-3. doi:10.1177/0009922812437930
- 14. Taylor L, Tan A, Coyle C, et al. Leveraging Social Determinants of Health: What Works? *PloS one*. August 17, 2016 2106;11(8):20. doi:10.1371/journal.pone.0160217
- 15. Shumway M, Boccellari A, O'Brien K, Okin RL. Cost-effectiveness of clinical case management for ED frequent users: results of a randomized trial. *The American journal of emergency medicine*. Feb 2008;26(2):155-64. doi:10.1016/j.ajem.2007.04.021
- 16. Berkowitz SA, Hulberg AC, Standish S, Reznor G, Atlas SJ. Addressing Unmet Basic Resource Needs as Part of Chronic Cardiometabolic Disease Management. *JAMA internal medicine*. Feb 1 2017;177(2):244-252. doi:10.1001/jamainternmed.2016.7691
- 17. Hsieh HF, Shannon SE. Three approaches to qualitative content analysis. *Qual Health Res.* Nov 2005;15(9):1277-88. doi:10.1177/1049732305276687
- 18. Boyatzis R. *Transforming Qualitative Information: Themaic Analysis and Code Development*. Sage Publications; 1998.
- 19. Miles M, Huberman A, Huberman M. *Qualitative data analysis: An expanded sourcebook*. Sage Publications; 1994.

- 20. Miller WR, Rollnick S. Ten things that motivational interviewing is not. *Behavioural and cognitive psychotherapy*. 2009;37(2):129-140.
- 21. Miller WR, Rollnick S. *Motivational interviewing: Preparing people for change, 2nd ed.* Motivational interviewing: Preparing people for change, 2nd ed. The Guilford Press; 2002:xx, 428-xx, 428.


# Appendix A: Description of the Intervention and Randomization Unmet Needs Screen:

Veterans (anticipated N=1760) will be screened for unmet needs (index screen) and those identified as having at least one unmet need (target N=880) will be randomized to one of three study arms and screened again 6-months later. We will use the sealed opaque envelope program to generate randomization. For the index screen, a study Research Assistant (RA) will administer the screening instrument to Veterans by phone prior to the Veteran's upcoming primary care (PC) clinic appointment to gather data on nine unmet needs (full screen in **Appendix I**). Six months after the index screen, the RA will re-screen each Veteran participant by phone. For each completed screen, we will provide Veterans \$15 for their time.

After the RA determines each participant is eligible (see Section 5.2. Recruitment Methods), randomization will occur by the RA opening sealed envelopes that reveal the treatment assignments (screening, awareness, or assistance). Envelopes will be opened for each participant in the order they are recruited. The RA will then inform the participant of their assignment.

#### **Resource Sheets:**

For Veterans in the Awareness and Assistance arms, the RA will provide (via U.S mail) Resource Sheets tailored to the unmet needs identified in the index screen. During the index screen (by phone), the RA will inform the Veteran that they will receive a Resource Sheet in the mail and mail the Resource Sheets to the Veteran within two days of the index screen. During the index screen, the RA will additionally ask the Veteran if they would also like to receive the Resource Sheets via email. For Veterans who respond affirmatively, the RA will send the Resource Sheets as an email attachment during the index screen phone call and offer to review its content with them. The email message will be sent via encrypted email and will not solicit reply. (Appendix G contains the phone script for this interaction, and Appendix P contains the Resource Sheet email text and the cover letter for mailing.)

For each of the nine unmet needs, following the approach used in the VISN 1 pilot and at our academic affiliate hospital (Boston Medical Center), a Resource Sheet will include the names of available resources within VA and/or the local community that can help address the identified need(s) and contact information (e.g., address, phone, website, email) and hours of operation. (See **Appendix O** 

for sample Resource Sheets currently used in VISN 1 unmet need screening and referral pilot).

Prior to study initiation, we will contact all organizations listed on the Resource Sheets to determine if they have current capacity for referrals generated from our study. Organizations without such capacity will be replaced with other organizations with capacity. Then, following practices for regular updating of resource information used by our colleagues and by national organizations addressing unmet needs (e.g., Health Leads, NowPow), RAs at each site and in consultation with local SW services will contact the programs listed on the Resource Sheets monthly, to update status for accepting referrals and contact information. RAs will track and record time spent maintaining the Resource Sheets to identify the resource demands of this component of the intervention for replication purposes.

# **Social Work-Supported Referrals**

In the Assistance arm, we will hire and train social workers (one per site) to support Veterans to connect with resources following a standard operating procedure informed by current VA SW practices. Following the index screen and provision of tailored Resource Sheets, the RA will offer and encourage Veterans in this arm to receive assistance from a SW. Veterans may choose to opt out, but if they assent, the RA will provide the Veteran with the name and phone number of the SW who will contact the Veteran within two business days of the index screen (making up to five attempts to reach the Veteran by phone). During this initial call, the SW will use a standardized bio-psychosocial assessment tool used by VA SW and proven motivational interviewing methods<sup>20, 21</sup> to uncover details of the Veteran's unmet needs, identify barriers to resolving the unmet needs, and develop an action plan for the Veteran including how to overcome the identified barriers. In addition, following VA SW practice, the SW will call the resource(s) to which the Veteran has been referred to inform them the Veteran will be coming for services. The SW will conduct initial follow-up by phone one week after the interview/action plan development, with planned subsequent phone outreach every two weeks for up to seven weeks. At each call and as needed (i.e., if Veteran has not yet connected to services), the SW will again employ motivational interviewing methods with the goal of re-affirming the action plan or modifying it as needed. The SW will track and record all Veteran encounters in a research data base, including time spent, challenges and best practices identified.


VA Central IRR
# Appendix B: Protocol for Warm Hand-Off to Veterans Crisis Line

## Taken from the Quantitative Workstream Handbook

For those with "Higher" or "Indeterminate Higher" Risk:

→Offer Veterans Crisis Line and warm hand-off (Refer to VCL Warm Hand-off Instructions Page (see last page)). Use the phone number: 585-393-7938 and DO NOT provide this number to Veterans.

- → If the Veteran declines warm hand-off to VCL, attempt to keep the Veteran on the phone while also contacting the Veterans

  Crisis Line the VHA Suicide Prevention Office at 

  VHASuicidePReventionOffice@va.gov.
- → If the caller disconnects before the transfer can be made, send email to the VHA Suicide Prevention Office at the above email address.
- → VCL will continue outreach attempts until the Veteran is reached or for one week, and will involve the Veteran's local Suicide Prevention Coordinator (SPC) as appropriate.

Interviewer Reads: You mentioned earlier that you have had thoughts about harming yourself. [OR for those who refuse to answer question(s): You seem hesitant to answer questions about possible self-harm.] I want to encourage you to talk with your doctor or mental health provider about these thoughts, and I will send a message to the Suicide Prevention Coordinator at your VA Medical Center mentioning that you have expressed these concerns. They may contact you to discuss these concerns further. In addition, I can transfer you to someone at the Veterans Crisis Line so that you can talk further right now with someone who is qualified to help you in this situation.

- → In the rare occurrence that the interviewer is concerned about imminent risk (i.e., caller has already hurt self/others or has immediate plan to harm self/others and has access to means to inflict harm), contact Veterans Crisis Line (VCL) for dispatch of emergency services by calling the VCL Warm Transfer number: 585-393-7938 (DO NOT provide this number to Veterans).
- → Provide Veteran information for Veterans Crisis Line: name, current location, phone number, date of birth

**Interviewer Reads (for VCL warm hand-off):** I am concerned for your safety and would like to reach out to the Veterans Crisis Line on your behalf. There will

be a brief silence, please hold on the line while I transfer you to someone who is qualified to help you.

Interviewer Reads (if Veteran refuses): I'd like to encourage you to contact your doctor or mental health provider and to call the Crisis Line whenever you need to. Their number is 1-800-273-TALK. Thank you for your time, and I wish you all the best with your continued treatment.

#### **Abbreviated Script**

Step 1: Once the Veteran has agreed to speak with someone at the VCL, let them know that there will be a brief silence as you get a VCL representative on the line.

Step 2: Press "Flash", "Flashlink" or "Conference" button depending on the type of phone you are using.

[Veteran will now be on hold]

Step 3: Dial the VCL direct line. (585-393-7938)

Step 4: Once the VCL representative is on the line, describe the situation and provide the Veteran's contact information

Step 5: Press "Flash", "Flashlink" or "Conference" to get the Veteran back on the line.

[At this point all three people will be present.]

Step 6: Let the Veteran know that you will be getting off the line and hang up.

#### **Additional Notes**

- Call VCL ahead of time as it takes a while to connect
- Connect to the direct line (1-800 #) only if a warm hand-off is wanted
- Email is great way to connect with the VCL if there is a disconnection or if the Veteran declined a warm hand-off
- Provide background information of the Veteran to the VLC including birthday, location, phone #
- Must send suicidality forms encrypted
- Give the Veteran the 1-800 # if they want to use it later
- If you hang up, the Veteran and the VCL are still connected (unless you have a cell phone)





#### TRANSFERRING A CALL TO THE VETERANS CRISIS LINE (VCL)

- Determine if the caller is in distress. Signs of Distress: a. Remain calm and listen. · Emotional (crying, loud, yelling) · Making concerning statements like: b. Ask the question: "Sometimes when people are (upset/angry/in pain/etc.) they think about - My family would be better off if I wasn't here. suicide. Are you thinking about killing yourself - I can't go on like this. or someone else?" - No one can help me. Route caller to YES appropriate local NOT suicidal, homicidal, or in crisis Suicidal, homicidal, or in crisis resources.
- Assess if caller is at imminent risk (has already hurt self/others or has immediate plan to harm self/others and has access to means).
  - a. Notify your supervisor (or other staff) of the situation.
  - b. Try to obtain Veteran's information (phone number, name, last four digits of Social Security number, location).
  - c. Have supervisor (or other staff) immediately contact 585-393-7938 for safety check.
  - d. Remain on the phone with caller until emergency personnel arrive.
- 3. If caller is not at imminent risk, collect information:
  - a. Caller's phone number (caller ID or ask for their phone number)
  - b. Veteran's name
  - c. Veteran's Social Security number (or last four digits of the SSN)
  - d. Veteran's current location
- 4. Transfer the call:
  - a. Explain that you will conference a VCL staff member into the call.
  - b. Call 1-800-273-8255, Press 1.
  - c. Complete a warm transfer: When the VCL responder answers, identify yourself and the office you are calling from. Explain what is going on and provide the information that you collected about the caller before bringing the caller on the line.
  - d. Inform caller that you will hang up and he or she is in good hands with the VCL responder.
  - e. Make sure the caller is on the call with the VCL responder before hanging up.
  - f. Document the initial call and warm transfer to VCL in a CPRS administrative progress note or Report of Contact (VA Form 119), as required locally. Notify your supervisor, per facility procedure or protocol.

For more information about the Veterans Crisis Line, visit **VeteransCrisisLine.net**For more information about VA's mental health resources, visit **www.mentalhealth.va.gov** 

© 7/15 VHA

# **Appendix C: Cover Letter Inviting Veteran Participation**

«letter\_date»

«FName» «LName»

«Address 1», «Address 2»

«City», «State», «Zip»

Dear «Salutation»,

The Veterans Health Administration (VHA) understands that health begins with where Veterans live and work. For this reason, a team of VHA researchers are doing a research study to identify Veterans' needs (things like not having enough food or difficulty paying utilities) and connect Veterans to resources that can address their needs. **We are writing to invite you to participate in this study**.

The study aims to understand how VHA can better meet the resource needs of Veterans. If you are interested in learning more, a researcher will contact you by telephone to explain the study and answer any questions you might have.

Your participation is completely voluntary. We sincerely hope that you will be willing to assist us in this effort. We need as many Veterans as possible to participate so the results of this study will be meaningful. Please read the enclosed **information sheet.** It provides more details about the study.

If you do not want us to contact you about this study, please return the enclosed **postcard** so we will know not to call you. However, if you are interested in learning more, you do not have to do anything. If we do not receive your postcard within the next week, a member of the research team may contact you to discuss the study.

If you have any questions, please contact the project manager at 857-364-2350. On behalf of the research team and those Veterans who may benefit from the results of the study, we thank you in advance for your help.

Sincerely,

Deborah Gurewich, PhD Study Lead

# **Appendix D: Study Fact Sheet**

#### STUDY FACT SHEET

**Study Title:** The Effects of Screening and Referral for Social Determinants of Health on Veterans' Outcomes

Name of Study Lead (also called "Principal Investigator"): Deborah Gurewich, PhD

Name of Study Lead at your VA (also call "Local Site Investigator"): (insert relevant name)

- **1. What is the purpose of the study?** To understand how the Veterans Health Administration (VHA) can best help Veterans who have *resource needs*. *Resource needs* are also called social determinants of health. These are things like having trouble paying for housing or a hard time paying important bills, like electric or gas bills.
- **2.Who is invited to participate?** You are eligible to participate if you
  - *a*) have heart disease or cardiovascular disease (CVD) or are at risk for heart disease (for example, because you have high blood pressure), *and*
  - b) get primary care at the Boston, Charleston, or Philadelphia VA Healthcare Systems.
- 3. What does the study involve and how long will it last? The study has two parts.

In **Part One**, someone from the research team will call you. They will want to talk for about 30 minutes. They will go over the study and answer any questions you might have. Next, they will conduct a brief questionnaire with you about your resource needs (for example, they will ask about your housing). Depending on your answers, you may be eligible for Part Two of the study. If you are not eligible for Part Two, that will be the end of your participation in the study.

If you are eligible for **Part Two** of the study, you will be contacted by phone two more times – eight weeks and six months after the first telephone call. During these calls, a researcher will conduct brief questionnaires with you about your resource needs. These phone calls should take only 5-10 minutes.

For Part Two of the study, you will be randomly assigned to one of three study groups: A, B, or C (see Table 1). Being randomly assigned is like a flip of a coin for which group you would be placed in.

- Group A: Participants in this group will receive a postcard listing local and national VHA help lines that may help with resource needs.
- Group B: Participants in this group will receive a postcard and also a written list of resources (i.e., agencies and programs) tailored to each participant's specific resource needs.
- Group C: Participants in this group will receive a postcard, a written list of resources, and also be offered help from a social worker who is part of the research team. The social worker may contact you by phone to learn more about your resource needs and help you connect to agencies and programs. The social worker could contact the you by phone up to 5 more times.

If you are in Groups B or C, you might also be asked to participate in a phone interview. In contrast to the brief questionnaires described above, the phone interview will involve a longer list of questions and will take more time, we estimate 45-60 minutes. If you are selected for an interview, a member of the research team will contact you by phone between months 7 and 12. If you agree, the researcher will then schedule a time that is convenient for you to conduct the interview. Before the interview begins, we will ask your permission to audio record the interview. If you do not want the interview recorded, that is Ok and you can still participate in the interview. During the interview you will be asked about your experience participating in the study. Veterans who participate in Part Two of study will be in the study for 12 months.

Table 1. What Participants Will Receive by Study Group

| Group A | Group B | Group C |
|---|---|---|
| Postcard listing local and national VHA help lines | <ul> <li>Postcard listing local and national VHA help lines</li> <li>Resource sheet listing agencies and programs to address specific resource needs</li> </ul> | <ul> <li>Postcard listing local and national VHA help lines</li> <li>Resource sheet listing agencies and programs to address specific resource needs</li> <li>Assistance from a Social Worker to help connect to agencies and programs</li> </ul> |

- **4. What are the benefits of participating?** People who participate in this study may have a better understanding of the resources that can help Veterans with resource needs. Your participation may also add much needed knowledge about resource needs among Veterans and how the VHA can better meet the needs of Veterans with resource needs.
- **5. What are the possible risks or discomforts of participating?** Some people may feel uncomfortable or upset discussing resource needs during the telephone calls with research staff. You may choose to skip a question or stop the telephone call at any time. You can also withdraw from the study at any time. Some people may find the telephone calls inconvenient. We will make every effort to schedule phone calls when it is convenient for you and will try to keep them short. Finally, there is a general risk of loss of confidentiality, but we believe this risk is minimal.
- **6.** How will my private information be protected and who will have access to it? Information collected for this research study will be kept confidential as required by law and will <u>not</u> be shared with your care team. However, you are welcome to follow-up with your care team at any time during your participation this the study. The results of this study may be published for scientific purposes, but your record or identity will not be revealed unless required by law. We will store your information in ways we think are secure. We will store paper files in locked cabinets. We will store electronic files in computer systems with password protection and encryption. However, we cannot guarantee complete confidentiality. To help protect your personal information, we will assign you a study ID so that your identifiable information is not connected to you.

We will limit access to your personal information to members of the research team who need to review this information in order to conduct the study. In addition, a description of this study will be available at <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a> as required by U.S law. This website will not include information that can identify you.

Your research records will be destroyed in accordance with the VHA Record Control Schedule (www1.va.gov/VHAPUBLICATIONS/RCS10/rcs10-1/pdf). Records will be destroyed when allowed in the following manner: Paper records will be shredded; electronic records and audio recordings will be destroyed in a manner in which they cannot be retrieved.

Participating in this study will not affect your VHA healthcare including your healthcare providers' ability to see your records as part of normal care and will not affect your right to have access to your records during and after the study is completed.

There are times when we might have to show your records to other people. For example, someone from the Office of Human Research Protections, the Government Accountability Office, the Office of the Inspector General, the VA Office of Research Oversight, the VA Central IRB, our local Research and Development Committee, and other study monitors may look at or copy portions of records that identify you.

- **7. What are the costs of participating in the study?** You will not be charged for any activities or procedures that are part of this study.
- **8.** Do I have to take part in this study? No. Participating in the study is voluntary and if you refuse to take part in the study, there will be no penalty or loss of benefits to which you are otherwise entitled to from the VHA. There are also no consequences if you decide to withdraw from the study. In this instance, for data already collected prior to your withdrawal, the research team may continue to review the data already collected for the study but will not collect further information from you.
- **9. Who do I contact about this study of I have questions?** If you have any questions about the research study, concerns or complaints, you may contact the project manager at 857-364-2350. If you have questions about your rights as a study participant, or want to make sure the study is valid, you may contact the VHA Central Institutional Review Board toll free at 1-877-254-3130. This is the Board that is responsible for overseeing the safety of human participants in this study. You may call them at (insert contact information) if you have questions, complaints or concerns about the study or if you would like to obtain information or offer input.
- **10. Will I be compensated for being in this study?** As a thank you for your participation, you will receive a \$15 payment for each brief questionnaire you complete and a \$25 payment if you participate in a telephone interview. The form of payment (for example, check/voucher, gift card, etc.) may vary depending on the VA in which you get your care.


43

# **Appendix E: Resource Postcards**





# Are you in need of assistance now?

VA Boston Healthcare System, Patient Call Center, 150 S. Huntington Ave, Jamaica Plain MA 02130: (857) 364-4418

VA Veterans Crisis Line: 1-800-273-8255 (Press 1)

National Call Center for Homeless Veterans: 1-877-4AID-VET (4243-838)





# Are you in need of assistance now?

**Ralph H. Johnson VA Medical Center,** 109 Bee Street, Charleston SC 29401: 843-577-5011 or 888-878-6884

VA Veterans Crisis Line: 1-800-273-8255 (Press 1)

44

National Call Center for Homeless Veterans: 1-877-4AID-VET (4243-838)


VA Central IRB Effective Date: November 29, 2022





# Are you in need of assistance now?

Crescenz VA Medical Center (3900 Woodland Ave, Philadelphia PA 19104): 215-823-5800 | 800-949-1001

VA Veterans Crisis Line: 1-800-273-8255 (Press 1)

45

National Call Center for Homeless Veterans: 1-877-4AID-VET (4243-838)


VA Central IRB
Effective Date: November 29, 2023

# Appendix F: Opt-Out (Do-not-contact) Postcard





# Thank you, but I do not wish to be contacted for this study.

[Participant ID number]

#### Mail to:

VA Center for Health Organization & Implementation Research Boston VA Medical Center Attn: Rory Ostrow 150 S. Huntington Avenue (152-M)

Boston, MA 02130

46

# **Appendix G: Veteran Recruitment Phone Script**

| P | h | n | n | е | C | n | n | ta | C | ŀ٠ |
|---|---|---|---|---|---|---|---|----|---|----|

<u>Not Present:</u> Hello, my name is\_\_\_\_\_\_, I'm calling from the [**Name of VAMC**]. I am trying to reach [**Name of Veteran**]. I'll call back another time, thank you. Is there a good time to try calling back?

**Voicemail:** Hello, my name is **[name of research team member]** and I work at the **[Name of VAMC]**. I wanted to speak with **[Name of Veteran]** about a letter we sent a few weeks ago regarding a research study. If you are interested in learning more about this study, please contact me at 781-687-**[extension]**. If you get my voicemail please leave your name, the best number to reach you at, and the most convenient times to reach you. Thank you.

<u>Present</u>: Hello, my name is [name of research team member] and I work at the [Name of VAMC]. I wanted to speak with you about a letter we sent you a few weeks ago about a research study.

1. Do you have a minute?

If Yes: We are conducting a research study about Veterans' resource needs. We sent you a letter a couple of weeks ago that included a Study Fact Sheet, describing the study. Do you remember getting it?

If Yes: (SKIP TO #2)

**If No:** I apologize for that. We can send you another letter if you would like. I can also tell you about the study now. Is that okay?

**No:** Okay, great. I will make sure a letter is sent to you. I just want to confirm your mailing address **[confirm]**. Thank you for your time. If I don't hear from you in 2 weeks I will call back and see if you are interested in participating. (*END CALL*)

Yes: (SKIP TO #3A)

**If No**: Ok, can I schedule another time to call you to describe the study and see if you might be interested in participating?

If Yes: (SCHEDULE A TIME)

If No: Thank you for your time. Good-bye.

2. Would you be interested in getting some more information about the study?

**If not Interested:** Thank you for your time. Good-bye.

If interested: (GO TO #3)

3. Ok great. Let me describe the study to you and what it means to participate. The letter you received included a Study Fact Sheet. Do you have the Fact Sheet?

**If YES**: Great, it would be helpful to have the Study Fact Sheet in front of you, so we can go through it together. I can wait while you get it. (WAIT AS NEEDED AND THEN GO TO #4)

If NO: No problem at all. (GO TO #3A)

- **3a**. I will read the information in the Fact Sheet to you, and you will have a chance to ask questions. Let me first tell you about the study aims:
  - (FOLLOW STUDY FACT SHEET #1 AND #2)
  - When done: Do you have any questions? (RESPOND TO ANY QUESTIONS ASKED)

**3b**. Now let me describe what it means to participate:

- (FOLLOW STUDY FACT SHEET #3, FIRST TWO PARAGRAPHS)
- When done with 2<sup>nd</sup> paragraph: Do you have any questions? (RESPOND TO ANY QUESTIONS ASKED)
- Does this sound like something you would like to do?

If Yes: (GO TO #3C)

If No: Thank you for your time today. Goodbye.

- **3c**. I am glad you are interested. There are a few more things we need to review before you agree to participate and enter the study:
  - (FOLLOW STUDY FACT SHEET #3, LAST TWO PARAGRAPHS)
  - When done: Do you have any questions? (RESPOND TO ANY OUESTIONS ASKED)
  - (FOLLOW STUDY FACT SHEET ITEM 4 THRU 9)
  - When done: Do you have any questions? (RESPOND TO ANY QUESTIONS ASKED)
  - (SKIP TO #5)
- 4. Since you have the Study Fact Sheet, I will review it with you in summary. Afterwards, you will have the opportunity to ask questions, and to confirm that you understand your role in the study. Does this sound OK? (ADDRESS ANY QUESTIONS AND PROCEED)
  - The purpose of the study is to identify the resource needs that Veterans have (things like not having enough food) and understand how VHA can best connect Veterans with services and programs that can address their needs. Your participation in the study would last for 12 months.

- The study involves two parts. In Part One, someone from the research team will call you to conduct a brief questionnaire about your resource needs. Depending on your answers, you may be eligible for Part Two of the study. If you are eligible for Part Two, a member of the research team will contact you by phone two more times to administer brief questionnaires about your resource needs. These phone calls should take only 5-10 minutes.
- For the second part of the study, you will be randomly assigned to one of three study groups (random is like a flip of a coin). Participants in different groups will receive varying levels of assistance in connecting to resources. This is detailed in Table 1 in the Fact Sheet.
- For the second part of the study, you may also be invited to participate in one 45-60 minute phone interview.

4a. Do you have any questions so far about what the study involves and how long it would last? (RESPOND TO ANY QUESTIONS ASKED)

- o There are a few key additional points I want to highlight from the Study Fact Sheet. These include:
  - This study involves research.
  - Your participation is completely voluntary and if you choose to participate, you can withdraw at any time.
  - If you do participate, the information we collect from you will be kept confidential and your identity will not be revealed in any of the results we report or publish.
  - The risks of participating are that you may get upset answering questions about resource needs or may find the phone calls inconvenient. We will do everything we can to minimize these risks. The benefit of participating is that you may have a better idea about available resources; you may also help VA in doing a better job serving Veterans.
  - There are no costs associated with participating in the study. As a thank you for participation, you will receive a \$15 gift card to CVS\* for each brief questionnaire you complete. And, if you're selected (and agree) to participate in an interview, you will receive a \$25 gift card.

\*(For CIRB: The nature of the participant payment varies by site. In Boston (prime site), participants will receive CVS gift cards; in Philadelphia, participants can receive a voucher/check or direct deposit; in Charleston, participants can receive payment via direct deposit or on a VA DirectExpress debit card. Each site has submitted a version of the Recruitment Phone Script that is tailored to their specific payment method. This version is for the prime site, Boston.)

4b. Do you have any questions? (RESPOND TO ANY QUESTIONS ASKED)

5. Do you agree to participate in the study?

If No: Thank you very much for your time today. Goodbye.

**If Yes:** Thank you for agreeing to participate in this study! We really appreciate it. *(ENTHUSIASTIC RESPONSE)* If you have time now, about 10 minutes, we can get started with Part One right now.

**If don't have time**: When is a good time for you to answer some questions about your resource needs? (SCHEDULE A TIME AND CONFIRM BEST CONTACT NUMBER)

If have time now: (GO TO #6)

- 6. Complete unmet need survey. (For CIRB: See Appendix I)
- 7. **Among participants who identified zero needs**: Thank you for completing Part One of the study. It appears that you are not eligible for Part Two of this study, so today's call will end the study team's contact with you. We will be mailing you a \$15 gift card\* for your participation. \*(<u>CIRB Note</u>: local site payment process differs across sites, as detailed in their respective CIRB amendments. This appendix is the Boston version.)

7a. Do you have any questions (RESPOND TO ANY QUESTIONS ASKED).

Thank so much you for your time (END CALL).

- 8. Among Participants who identified one or more needs, randomize to one of three study arms.
- 9. Among participants randomized to Arm 1 (Screening): Thank you for completing Part One of the study. You are eligible for Part Two of the study and have been randomized to Group A. This means that in 8 weeks, I will recontact you to ask a few more questions about your needs. Do you have any questions? (RESPOND TO ANY QUESTIONS ASKED) (MENTION GIFT CARD AND VERIFY MAILING ADDRESS\*.) Thank you for your time.
- \*(<u>CIRB Note</u>: local sites will explain their payment process, which differs from the prime site)
- 10. Among participants randomized to Arm 2 (Awareness): Thank you for completing Part One of the study. You are eligible for Part Two of the study and have been randomized to Group B. I would like to provide you with some written material about programs and agencies that might be able to help you with the needs you identified. I will mail you this material within the next two business days. If you like, I can also email the material to you right now and we can review it together over the phone. Would you like to do that?

**If Yes to email**: Great, I can email that to you right now. (CONFIRM/ASK FOR PARTICIPANT'S EMAIL ADDRESS AND SEND ENCRYPTED EMAIL.)

If No to email: No problem. You can look for a written list of resources in the mail in the next several days. The information will include my phone number in case you have any questions about the information once you receive it.

10a. I will also be mailing you a \$15 gift card\* to thank you for your time. And in 8 weeks, I will recontact you to ask a few more questions about your needs. Do you have any questions? (RESPOND TO ANY QUESTIONS ASKED) (VERIFY MAILING ADDRESS FOR GIFT CARD)\* Thank you for your time.

\*(<u>CIRB Note</u>: local sites will explain their payment process, which differs from the prime site.)

11. Among participants randomized to Arm 3 (Assistance): Thank you for completing Part One of the study. You are eligible for Part Two of the study and have been randomized to Group C. I would like to provide you with some written material about programs and agencies that might be able to help you with the needs you identified. I will mail you this material within the next two business days. If you like, I can also email the material to you right now and we can review it together over the phone. Would you like to do that?

If Yes to email: Great, I can email that to you right now. (CONFIRM/ASK FOR PARTICIPANT'S EMAIL ADDRESS AND SEND ENCRYPTED EMAIL.)

If No: to email: No problem. You can look for a written list of resources in the mail in the next several days. The information will include my phone number in case you have any questions about the information once you receive it.

11a. I would also like offer you the assistance of a Social Worker (SW), who can assist you to connect to programs and agencies that might be able to help with the needs you identified. Would you like to receive this assistance?

**If No:** I encourage you to accept this assistance because it can be helpful. Are you sure you don't want assistance from a SW who can assist you to connect to services?

If does not want SW assistance: (GO TO #11b)

If wants SW assistance: (GO TO NEXT QUESTION)

If Yes: Terrific. The SW on the study team – his/her name is (insert name) -- will call you within two business days. Let me give you the name and number of the social worker so you have it. Do you have a pen and paper? (WAIT FOR PEN AND PAPER AND THEN PROVIDE NAME AND NUMBER)

11b. In 8 weeks, I will recontact you to ask a few more questions about your needs. Do you have any questions? (RESPOND TO ANY QUESTIONS ASKED) (MENTION GIFT CARD AND VERIFY MAILING ADDRESS)\* Thank you for your time.

\*(<u>CIRB Note</u>: local sites will explain their payment process, which differs from the prime site.)


52

# **Appendix H: Resource Representative Invitation Email**

Dear [Resource Representative Name],

A team of Veterans Health Administration (VHA) researchers are doing a research study to identify Veterans' needs (i.e., food insecurity, social isolation) and determine how the VHA can best connect Veterans to resources. We are writing to **invite your participation in our study**. **If you are interested in learning more, please reply to this email.** 

[Insert name of agency/VHA program] is among the resources that we have referred some of the Veterans participating in the study. Part of our study includes phone interviews with resource providers such as yours to learn more about providing services to Veterans. We anticipate the call will take about 30 minutes. It will be scheduled at a time convenient for you.

Your participation in this research study is completely voluntary. The interview data will be kept completely confidential. We will store the interview data in ways we think are secure – written materials will be stored in locked cabinets, and electronic material will be stored on secured, access-only servers. Your name nor the name of your Agency will not be shared in any presentations, reports, or papers summarizing our findings.

If you have any questions about our study or this invitation, please contact me at [phone #] or [email].

We sincerely hope you will be willing to assist us in this effort. The perspective of community agencies/VHA departments is critical to ensuring that VHA can address Veterans' resource needs.

We look forward to hearing from you. If we don't hear back from you in one week, we will follow-up again by email.

Sincerely,

[Site LSI Name]

[VAMC Name, Location]

53

# **Appendix I: Index Unmet Needs Screening Tool**

#### **DEMOGRAPHICS**

- 1. Please indicate which of following types of people currently live with you in your household (*check all that apply*)
  - My spouse or partner
  - My child(ren) under age 18
  - My adult child(ren) age 18 or older
  - My parent(s)
  - Extended family
  - Roommate(s) not related to me
  - Other individuals
- 2. Overall, which one of the following best describes how well you are managing financially these days?
  - Living comfortably
  - Doing OK
  - Just getting by
  - Finding it difficult to get by
- 3. Are you of Hispanic or Latino origin or descent?
  - Yes, Hispanic or Latino
  - No, not Hispanic or Latino
- 4. What is your race? Please select all that apply.
  - White
  - Black or African-American
  - Asian
  - Native Hawaiian or other Pacific Islander
  - American Indian or Alaska Native
  - Other
- 5. What is your gender
  - Man
  - Woman
  - Transgender man
  - Transgender woman
  - Non-binary
  - Other

#### **HOUSING AND UTILITIES**

- 6. In the past 6 months, have you been living in stable housing that you own, rent, or stay in as part of a household?
  - Yes
  - No

- 7. Are you worried or concerned that in the next 2 months you may NOT have stable housing that you own, rent, or stay in as part of a household?
  - Yes
  - No
    - 7a. (If Yes to Q6 or Q7): Are you already receiving assistance with your housing needs?
    - 7b. (If Yes to 7a): Would you like additional assistance?
    - 7c. (If No to 7a): Would you like assistance with your housing needs?
- 8. In the past 6 months has the electric, gas, oil or water company threatened to shut off service in your home?
  - Yes
  - No
  - · Already shut off
  - Not applicable
    - 8a. (If Yes/Already shut off): Are you already receiving assistance with your gas, oil or water company needs?
    - 8b. (If Yes to 8a): Would you like additional assistance?
    - 8c. (If No to 8a): Would you like assistance with your gas, oil or water company needs?

#### **EMPLOYMENT AND FOOD**

- 9. Are you currently:
  - Employed for wages
  - Self-employed
  - Out of work for 1 year or more
  - Out of work for less than 1 year
  - A Homemaker
  - A Student
  - Retired
  - Unable to work
    - 9a. Do you want help finding or keeping work or a job (check all that apply)?
      - Yes, help finding a job
      - Yes, help keeping work
      - I do not want or need help
      - I am already receiving assistance with my employment needs
- 10. How often were the following statements true for you in the past 6 months?
  - i. Within the past 6 months, you worried that your food would run out before you got money to buy more.
    - Often true
    - Sometimes true

Never true

ii. Within the past 6 months, the food you bought just didn't last and you didn't have money to get more.

- Often true
- Sometimes true
- Never true

10a. (If Often/Sometimes true to 10i or10ii): Are you already receiving assistance with your food needs?

10b. (If Yes to 10a): Would you like additional assistance?

10c. (If No to 10a): Would you like assistance with your food needs?

#### **LEGAL AND TRANSPORTATION**

- 11. Are you currently dealing with any legal issues, for which you may need assistance?
  - Yes
  - No
    - 11a. (If Yes): Are you already receiving assistance with your legal needs?
    - 11b. (If Yes to 11a): Would you like additional assistance?
    - 11c. (If No to 11a): Would you like assistance with your legal needs?
- 12. In the past 6 months, has lack of transportation kept you from medical appointments, meetings, work, or getting things needed for daily living: *Check all that apply* 
  - Yes, it has kept me from medical appointments or from getting my medications
  - Yes, it has kept me from non-medical meetings, appointments, or getting the things that I need
  - No
    - 12a. (If Yes): Are you already receiving assistance with your transportation needs?
    - 12b. (If Yes to 12a): Would you like additional assistance?
    - 12c. (If No to 12a): Would you like assistance with your transportation needs?

## SOCIAL AND EMOTIONAL STATUS

- 13. In the last 6 months, how often did you feel lonely or isolated?
  - Never
  - Rarely
  - Sometimes
  - Often

- Always
  - 13a. (If Sometimes/Often/Always): Are you already receiving assistance with your feelings of loneliness or isolation?
  - 13b. (If Yes to 13a): Would you like additional assistance?
  - 13c. (If No to 13a): Would you like assistance with your feelings of loneliness or isolation?
- 14. Stress is when someone feels tense, nervous, anxious, or can't sleep at night because their mind is troubled. In the last 6 months, how often did you feel stressed?
  - Not at all
  - A little bit
  - Somewhat
  - Quite a bit
  - Very much
    - 14a. (If Somewhat/Quite a bit/Very much): Are you already receiving assistance with your feelings of stress?
    - 14b. (If Yes to 14a): Would you like additional assistance?
    - 14c. (If No to 14a): Would you like assistance with your feelings of stress?

#### **EXPOSURE TO VIOLENCE**

- 15. Is anyone in your life hurting or threatening you?
  - Yes
  - No
  - 15a. (If Sometimes/Often/Always): Are you already receiving assistance with your being hurt or threatened?
  - 15b. (If Yes to 15a): Would you like additional assistance?

57

15c. (If No to 15a): Would you like assistance with your being hurt or threatened?

# **Appendix J: Eight-Week Follow-Up Survey**

| | g |
|---|---|
| Phone Contac | : <u>t:</u> |
| Hello, my name<br>reach <b>[Name o</b> | e is, I'm calling from the ( <b>Name of VAMC</b> ). I am trying to of <b>Veteran</b> ]. |
| Not Present:<br>back? | I'll call back another time, thank you. Is there a good time to try calling |
| (Name of VAM<br>Needs Study. I<br>study, it will on<br>[extension]. If | llo, my name is <b>[name of research team member]</b> , I am calling from the <b>IC</b> ). I wanted to speak with <b>[Name of Veteran]</b> about the Resource t's time to complete one of the brief questionnaires that are part of this ly take about 5 minutes to complete. Please contact me at 781-687-you get my voicemail please leave your name, the best number to reach most convenient times to reach you. Thank you. |
| (Name of VAM participating in. | my names is <b>[name of research team member]</b> and I work at the <b>IC)</b> . I wanted to speak with you about the Resource Needs Study you are It's time to complete one of the brief questionnaires that are part of this ly take about 5 minutes to complete. Do you have a few minutes now? |
| | When is a good time for you to answer some questions about your social stances? (SCHEDULE A TIME AND CONFIRM BEST CONTACT ER) |
| If Yes: | Great, let's get started. |
| Screening Sur | rvey |
| any new progra<br>Yes | st talked on [insert index screening date], were you able to connect with ams or services for help with [insert needs identified from index screen)? to Q5) |
| 2. Which progr | ams or services did you connect with? |
| 3. Were you ab<br>Yes<br>No | ole to get the help you wanted from this (these) program(s)? |
| 4. How did you<br>Probes<br>phone o<br>walk in<br>web-ba | |

58 *Version: 11/06/2023* 

e-mail




59

VA Central IRB Effective Date: November 29, 2023

# Appendix K: Six-Month Follow-Up Survey

| Phone Contact: | | |
|---|---|---|
| Hello, my name is<br>reach [Name of Veteran]. | _, I'm calling from the ( <b>Name of VAMC</b> ). | I am trying to |

**Not Present:** I'll call back another time, thank you. Is there a good time to try calling back?

<u>Voicemail:</u> Hello, my name is [name of research team member], I am calling from the (Name of VAMC). I wanted to speak with [Name of Veteran] about the Resource Needs Study. It's time to complete one of the brief questionnaires that are part of this study, it will only take about 10 minutes to complete. Please contact me at 781-687-[extension]. If you get my voicemail please leave your name, the best number to reach you at, and the most convenient times to reach you. Thank you.

<u>Present</u>: Hello, my names is [name of research team member] and I work at the (Name of VAMC). I wanted to speak with you about the Resource Needs Study you are participating in. It's time to complete one of the brief questionnaires that are part of this study, it will only take about 10 minutes to complete. Do you have a few minutes now?

**If No**: When is a good time for you to answer some questions about your social circumstances? (SCHEDULE A TIME AND CONFIRM BEST CONTACT NUMBER)

If Yes: Great, let's get started.

#### Screening Survey

#### **HOUSING AND UTILITIES**

- 1. In the past 6 months, have you been living in stable housing that you own, rent, or stay in as part of a household?
  - Yes
  - No
- 2. Are you worried or concerned that in the next 2 months you may NOT have stable housing that you own, rent, or stay in as part of a household?
  - Yes
  - No
- 3. In the past 6 months has the electric, gas, oil or water company threatened to shut off service in your home?
  - Yes
  - No
  - Already shut off
  - Not applicable

#### **EMPLOYMENT AND FOOD**

- 4. Are you currently:
  - Employed for wages
  - Self-employed
  - Out of work for 1 year or more
  - Out of work for less than 1 year
  - A Homemaker
  - A Student
  - Retired
  - Unable to work
- 5. How often were the following statements true for you in the past 6 months?
  - i. Within the past 6 months, you worried that your food would run out before you got money to buy more.
    - Often true
    - Sometimes true
    - Never true
  - ii. Within the past 6 months, the food you bought just didn't last and you didn't have money to get more.
    - Often true
    - Sometimes true
    - Never true

#### **LEGAL AND TRANSPORTATION**

- 6. Are you currently dealing with any legal issues, for which you may need assistance?
  - Yes
  - No
- 7. In the past 6 months, has lack of transportation kept you from medical appointments, meetings, work, or getting things needed for daily living: Check all that apply
  - Yes, it has kept me from medical appointments or from getting my medications
  - Yes, it has kept me from non-medical meetings, appointments, or getting the things that I need
  - No

#### **SOCIAL AND EMOTIONAL STATUS**

- 8. In the last 6 months, how often did you feel lonely or isolated?
  - Never
  - Rarely
  - Sometimes
  - Often
  - Always

- 9. Stress is when someone feels tense, nervous, anxious, or can't sleep at night because their mind is troubled. In the last 6 months, how often did you feel stressed?
  - Not at all
  - A little bit
  - Somewhat
  - Quite a bit
  - Very much

## **EXPOSURE TO VIOLENCE**

- 10. Is anyone in your life hurting or threatening you?
  - Yes
  - No


62

# **Appendix L: Veteran Interview Guide (Not Connected)**

#### **Phone Script**

Hello, my name is **[RA's name]** from **[name of VAMC]**. I'm calling to talk to you about the Resource Needs Study you are participating in.

As a participant in our study, you recently completed a questionnaire and indicated that you had the following needs [insert domain(s)].

I'd like to ask you a few questions about this/these need(s), as well as your experience participating in our study. This should take about [30-45 minutes depending on how much you have to say].

Do you have time to talk now, or would you like to schedule another time?

#### If scheduling for later:

OK, sure, when is a good time for us to call you for this interview? (CONFIRM DATE/TIME)

Is this the best number to reach you at that time? (CONFIRM PHONE NUMBER)

Thank you for you participating, I look forward to talking with you at **(agreed date/time).** 

#### If interviewing now:

Great, thank you!

(Informed Consent Reminder) Before we begin, I want to remind you that you are participating in research; your participation is voluntary; and you may decline to answer any of my questions or stop this interview at any time. I would like to use an audio-recorder so I can do a good job of listening to you. Is that alright with you?

Remember that we will not use your name or identify you in any way in presentations

Do you have any questions before we begin? (RESPOND TO ANY QUESTIONS)

Do you have any questions before I turn on the audio recorder? (RESPOND TO ANY QUESTIONS)

OK, let's get started. (TURN ON AUDIO RECORDER, IF RESPONDENT AGREED)

#### Interview Guide

Note: This is a semi-structured, qualitative interview guide meant to be used flexibly. The interviewer may follow-up with further open-ended questions and requests for clarification. The interviewer may also follow-up on issues raised by the participant. Questions may be asked in a different order, depending on the flow of conversation. Not all questions will be asked of each interviewee, as some questions may not be relevant to all subjects. [sub-questions are prompts]

- 1. To begin, it would be helpful for me to know a little about. Can you briefly tell me a little about yourself, like where you work, live or, who you live with?
- 2. Now let's talk about your experience participating in our study. As part of the study, you completed a questionnaire over the phone about your unmet needs (like whether you had reliable transportation) and whether you wanted assistance with the needs you have.
  - a. How did you experience that?
  - b. What did you like and not like?
  - c. What suggestions to you have about how VA could best learn about the resource needs that Veterans have?
- 3. In the questionnaire you indicated that you had the following needs [insert domains(s)]. I'd like to ask you a few questions about this/these need(s). And at any point, It would be helpful if you could make any important distinctions across before the pandemic, during the pandemic and now.
  - a. Tell me about your experience with [insert unmet need domain(s)], how long you have had this/these needs, how much you worry about this/these needs.
- 4. How did you feel about receiving a list of services and contact information that could help you to address your need(s) for [insert domain(s)]?
  - a. What worked for you about the experience?
  - b. What didn't work for you?
  - c. Are there ways these handouts could have been made more useful for you?
- 5. SW ARM ONLY How did you feel about a social worker assisting you to connect to services that might help you with your need for [insert domain(s)]?
  - a. What worked for you about the experience?
  - b. What didn't work for you?
  - c. Are there things the social worker could have done to be more helpful for you?
- 6. Among all the things that you need to manage in your life, how does [insert domain] need fit in?
- 7. (For respondents who tried but were unable to connect to new services) Through your participation in the study, we understand that you tried to connect with new services from (insert name(s) of program(s)/organization(s) but were unable to. Can you tell us about this experience?

- 8. (For respondents who did not try to connect to new services) Through your participation in the study, we understand that you did not try to connect with new services from (insert name(s) of program(s)/organization(s) Thinking back to when you were provided a list of services that might be able to help you with your needs and (if applicable) contacted by social worker to assist you in accessing services what were some of the reasons you didn't try to use these services?
- 9. What would have made it easier to connect with these services?
  - a. Probe:
  - b. Location
  - c. Access to phone and/or internet
  - d. Perceived ability to navigate social service delivery system
  - e. Assistance from others
- 10. In the thinking about your need(s) for [insert domain(s)], were you confident that available services within the VA or the community in which you live could help you with this/these need(s)? Why or why not?
- 11. Is there anything else you'd like to tell us about your experience participating in the study?


65

VA Central IRB

# **Appendix M: Veteran Interview Guide (Connected)**

#### **Phone Script**

Hello, my name is **[RA's name]** from **[name of VAMC]**. I'm calling to talk to you about the Resource Needs Study you are participating in.

As a participant in our study, you recently completed a questionnaire and indicated that you had the following needs [insert domain(s)].

I'd like to ask you a few questions about this/these need(s), as well as your experience participating in our study. This should take about 30-45 minutes depending on how much you have to say.

Do you have time to talk now, or would you like to schedule another time?

#### If scheduling for later:

OK, sure, when is a good time for us to call you for this interview? (CONFIRM DATE/TIME)

Is this the best number to reach you at that time? (CONFIRM PHONE NUMBER)

Thank you for you participating, I look forward to talking with you at **(agreed date/time).** 

#### If interviewing now:

Great, thank you!

(Informed Consent Reminder) Before we begin, I want to remind you that you are participating in research; your participation is voluntary; and you may decline to answer any of my questions or stop this interview at any time.

Remember that we will not use your name or identify you in any way in presentations of our study results. I would like to use an audio-recorder so I can do a good job of listening to you. Are you Ok with that?

Do you have any questions before we begin? (RESPOND TO ANY QUESTIONS)

OK, let's get started. (TURN ON AUDIO RECORDER, IF RESPONDENT AGREED)

#### Interview Guide

Note: This is a semi-structured, qualitative interview guide meant to be used flexibly. The interviewer may follow-up with further open-ended questions and requests for clarification. The interviewer may also follow-up on issues raised by the participant.

Questions may be asked in a different order, depending on the flow of conversation. Not all questions will be asked of each interviewee, as some questions may not be relevant to all subjects. [sub-questions are prompts]

- 1. To begin, it would be helpful for me to know a little about. Can you briefly tell me a little about yourself, like where you work, live or, who you live with.
- 2. Now let's talk about your experience participating in our study. As part of the study, you completed a questionnaire over the phone about your unmet needs (like whether you had reliable transportation) and whether you wanted assistance with the needs you have. How did you experience that? What did you like and not like about the experience? What suggestions do you have about how the VA could best learn about the resource needs Veterans have?
- 3. In the questionnaire you indicated that you had the following needs [insert domains(s)]. I'd like to ask you a few questions about this/these need(s). And at any point, It would be helpful if you could make any important distinctions across before the pandemic, during the pandemic and now.
  - a. Tell me about your experience with [insert unmet need domain(s)], how long you have had this/these needs, how much you worry about this/these needs.
- 4. How did you feel about receiving a list of services and contact information that could help you to address your need(s) for [insert domain(s)]?
  - a. What worked for you about the experience?
  - b. What didn't work for you?
  - c. Are there ways these handouts could have been made more useful for you?
- 5. SW ARM ONLY How did you feel about a social worker assisting you to connect to services that might help you with your need for [insert domain(s)]?
  - a. What worked for you about the experience?
  - b. What didn't work for you?
  - c. Are there things the social worker could have done to be more helpful for you?
- 6. Through your participation in the study, we understand that you received new services from [insert name(s) of program(s)/organization(s)].
  - a. Can you tell us a little about that?
  - b. Can you walk us through the steps you took to get these services? Was it easy to connect to these services? Why or why not? *Probes:* 
    - i. Location
    - ii. Access to phone and/or internet
    - iii. Perceived ability to navigate social service delivery system
    - iv. Assistance from others
  - c. What did you think about the organization[s] you were told about?
- 7. How was your experience receiving services?
  - a. How helpful was/were the service(s) in addressing your need(s)?
  - b. Are there things that worked well or did not?
  - c. How could the service(s) better meet your needs?

- d. What else should I know about the services you received?
- e. How could the VA better address your unmet needs? (probe for what would be most helpful for the respondent).
- 8. What did you think about the organization[s] you were told about?
- 9. Among all the things that you need to manage in your life, how does [insert domain] need fit in?
- 10. Is there anything else you'd like to tell us about you? Your experience participating in the study?


68

VA Central IRB Effective Date: November 29, 2023

# **Appendix N: Resource Representative Interview Guide**

#### Phone Script

Hello, my name is [RA Name] from [VAMC Name].

I'm calling to conduct an interview with you about your experience as a resource provider for the Veterans in our study identifying unmet resource needs.

Is this still a good time to talk?

**If No:** No problem, when will be a good time for us to talk? (ANSWER ANY QUESTIONS AND RESCHEDULE THE CALL.)

Great. I look forward to talking to you then.

If Yes: Great! This call should take about 30 minutes.

I want to remind you of a few things before we begin: your participation is completely voluntary; you can stop the interview at any time, and you may choose not to answer any question you are uncomfortable answering. Your answers will be kept completely confidential and we will not use your name to identify you in any results. I would like to use an audio-recorder so I can do a good job of listening to you. Are you Ok with that?

Do you have any questions before we begin? (ANSWER ANY QUESTIONS)

OK, let's get started. (TURN ON AUDIO RECORDER, IF RESPONDENT AGREED)

#### Interview Guide

Note: This is a semi-structured, qualitative interview guide meant to be used flexibly. The interviewer may follow-up with further open-ended questions and requests for clarification. The interviewer may also follow-up on issues raised by the participant. Questions may be asked in a different order, depending on the flow of conversation. Not all questions will be asked of each interviewee, as some questions may not be relevant to all subjects. [sub-questions are prompts]

- 1. Tell me a little about your work in general.
  - a. What specifically is your role?
- 2. Can you tell me about your program?
  - a. What kind of services does your program provide?
  - b. (For community-based programs): Can you tell me a little about your organization's relationship with the VA?
- 3. How do clients/patients typically find you?
  - a. Who is eligible for your program (inclusion and exclusion criteria)?

- b. (For VA programs): What types of VA providers/departments refer to you?
- c. (For community-based programs): What types of organizations, if any, refer to you?
- d. (For community-based programs only) Do you have a way of knowing if clients are Veterans?
- e. How could the referral process for your services be improved?
- 4. Can you tell me about the ebbs & flows in your work?
  - a. In particular, what about volume in utilization of your services?
  - b. During the past year, did you notice increased Veteran referrals to your programs and if so, how did you manage the uptick in referrals?
  - c. It would be helpful if you could make any important distinctions across before the pandemic, during the pandemic and now.
- 5. How does the potential for increased Veteran referrals for your services sit with you? What might you need to address an increase? What should VA know?
- 6. (For community-based programs only) Is there anything particular to Veterans when thinking about the services you provide and if so, please tell us about it.
- 7. (For community-based programs only) What does the VA need to know about working with your organization?
- 8. There is increasing incentivization for health care organizations like the VA to screen for unmet social needs and refer patients with identified needs to programs/organizations such as yours. What are your thoughts on this?
- 9. Is there anything else you'd like to share about how the VA can best address the unmet social needs of the Veterans they serve?
- 10. Given everything we've talked about today, is there anything else I should know? Something you thought I'd asked but didn't?

Thank you for your time.

# **Appendix O: Example Resource Sheets**

(See pages following)

#### Social Risk Factors Resource Guide: TRANSPORTATION RESOURCES

If you have any questions about the information provided below or want additional assistance contacting the programs, please contact Timothy Driscoll, 781-687-2374, Health Care for Homeless Veterans Program at Bedford VA.

**The Bedford Shuttle Services**: Shuttle service to Boston VA facilities and Bedford CBOC locations. You must be scheduled to utilize so please call (781) 687-2505 with questions. Seating is limited to scheduled Veterans. Full Listing of shuttle services and times and location of departure available [website will be provided here].

#### MBTA Cards, Social Work Service 781-687-2375

MBTA cards for Veteran's who are without funds and in need of transportation within the Mass Transit system.

**The Ride** is the T's Paratransit program, provides door-to door transportation to eligible people who cannot use general public transportation all or some of the time, because of a physical, cognitive or mental disability In order to use THE RIDE you must complete and submit an application. Per ADA regulations, 21 days is allowed to process applications upon receipt. Only completed signed original applications, mailed to the address below, will be considered for review. You will receive written notification of eligibility via U.S. mail.

[website for MBTA will be provided here]. MBTA Office for Transportation Access 10 Park Plaza - Room 5750 Boston, MA 02116 (800) 533-6282 in-state toll free (617) 222-5123 TTY (617) 222-5415

#### **Regional Transit Authority Contact Information**

72

You can learn more about regional or local transportation service options below:

CATA - Cape Ann Transportation Authority [website will be provided here] Gloucester (978) 283-7916

LRTA - Lowell Regional Transit Authority [website will be provided here] Lowell (978) 459-0164 TTY (800) 439-2370

**MWRTA - MetroWest Regional Transit Authority** [website will be provided here] **Framingham (508) 935-2222 1-888-996-9782** 

MVRTA - Merrimack Valley Regional Transit Authority [website will be provided here] Haverhill (978) 469-1254 (V/TTY)


VA Central IRB Effective Date: November 29, 2023

#### Social Risk Factors Resource Guide: FOOD SECURITY RESOURCES

If you have any questions about the information provided below or want additional assistance contacting the programs, please contact Timothy Driscoll, 781-687-2374, Health Care for Homeless Veterans Program at Bedford VA.

SNAP: Supplemental Nutrition Assistance Program – formerly known as SNAP. [website for SNAP will be provided here]

SNAP benefits are provided by the federal government and administered by DTA. Residents of the Commonwealth who participate in SNAP are families with children. elders and disabled. To apply for SNAP benefits, you may fill out the SNAP application to see if you are eligible to receive benefits. To find the Transitional Assistance office that covers your city/town, visit the above link and click on the "Transitional Assistance Office" link. If you are not sure which office to contact or you have questions about how to apply for DTA programs, please contact the DTA Application Information Hotline at 1-800-249-2007, Monday through Friday from 8:45 AM – 5:00 PM.

#### Some Local offices include:

#### Lawrence

15 Union Street Lawrence, MA 01840 Phone: (978) 725-7100 Fax: (978) 681-6216 Mon - Fri 7:00am to 5:00pm

#### Lowell

131 Davidson Street Lowell. MA 01852 Phone: (978) 446-2400 Fax: (978) 458-7563 Mon - Fri 7:00am to 5:00pm Fax: (617) 727-4567 Mon - Fri

7:00am to 5:00pm

#### To find a food pantry or free meal program near you, call:

The FoodSource Hotline Telephone: 1-800-645-8333 TTY: 1-800-377-1292

Web site: The FoodSource Hotline

Malden. MA 02148 Phone: (781) 388-7300 Fax: (617) 727-7493 Mon - Fri

7:45am to 5:00pm

Revere 300 Ocean Avenue Revere, MA 02151

200 Pleasant Street

Malden

Phone: (781) 286-7800 (800) 650-2560

Merrimack Valley Food Bank (Lowell)

Web site: Merrimack Valley Food Bank

Telephone: 978-454-7272

Greater Boston Food Bank (Eastern Massachusetts)

Telephone: 617-427-5200

Web site: The Greater Boston Food Bank - Get Help

#### Social Risk Factors Resource Guide: UTILITY ASSISTANCE RESOURCES

If you have any questions about the information provided below or want additional assistance contacting the programs, please contact Timothy Driscoll, 781-687-2374, Health Care for Homeless Veterans Program at Bedford VA.

Fuel Assistance: even if heat is included in your rent you may still be eligible for fuel assistance benefits as long as you are paying at least 30% of your gross income towards your rental portion. Fuel Assistance is open from November 1<sup>st</sup> to April 30<sup>th</sup>. Documentation needed includes: A.) Four most recent consecutive pay stubs from date of application or a letter from your employer indicating gross wages for the same time period. B.) Social Security numbers of everyone living in the household. C.) Proof of residency such as a rent receipt or real estate tax bill. D.) Utility bills including gas, electric, oil, wood, coal, propane or other. E.) There may be additional required documentation depending on family circumstances, living arrangements, or heating source.

Lawrence: 978.681.4900 Lowell: 978.459.6161 Haverhill: 978.373.1971 Bedford: 978.459.6161 Arlington: 781.643.2358

Individuals and families eligible for Fuel Assistance are automatically submitted to utility companies for enrollment in special discount programs.

- ☑ Low Income Gas Rate, sponsored by Bay State Gas, provides a discount of approximately 20% off their gas bill.
- Assurance phone for free phone to qualifying households
- ☑ Lifeline Telephone Assistance, sponsored by NYNEX, provides for a discount of \$9.50 on their telephone bill. Only one telephone line per household is eligible.
- ✓ Low income electric rate, R-2 rate, for Mass. Electric. This is a discounted rate of 33% off electric bills.
- ☑ Bay State Gas discounted Low Income Gas Rate [website will be provided here]
- Lifeline Telephone Assistance [website will be provided here] **SafeLink** Wireless Phone [website will be provided here]
- ☑ National Grid Discount Rate (R2 Rate) 1.800. 322-3223 and [website will be provided here]
- ☑ NSTAR (R2 Rate) 800-566-2080 or apply on line

#### Social Risk Factors Resource Guide: HOUSING STABILITY RESOURCES

If you have any questions about the information provided below or want additional assistance contacting the programs, please contact Timothy Driscoll, 781-687-2374, Health Care for Homeless Veterans Program at Bedford VA.

## HUD/VASH Program, Ed Fleming, Program Manager, 781-687-3521

Provide permanent housing options to homeless Veterans or Veterans at risk of homelessness as well as clinic case management support.

Healthcare for Homeless Veterans, Tim Driscoll, Program Manager 781-687-2374

Daily Walk-In Clinics to assist homeless Veterans. Provide clinical support to homeless Veterans around medical, mental health and substance use issues.

#### **FURNITURE RESOURCES**

| Household Goods Recycling of Massachusetts (978) 635-1710 | 530 Main<br>St. | Acton | MA | 01720 | HGRM<br>Particular Particular Politics |
|---|---|---|---|---|---|
| Project Home<br>Again<br>(978) 470-1356 | | Andover | MA | 01810 | projecthomeagain |
| My Brother's<br>Keeper<br>(508) 238-7512 | P.O. Box<br>338 | Easton | MA | 02356 | MY BROTHER'S KEEPER A State Class State on patter Section State State on patter Section State State on patter Section State State State on patter Section State St |
| Massachusetts Coalition for the Homeless (781) 595-7570 | 15 Bubier<br>St. | Lynn<br>(Boston) | MA | 01901 | BEADLAY 19 |
| Mission of<br>Deeds<br>(781) 944-9797 | 6 Chapin<br>Ave | Reading<br>(Boston) | MA | 01867 | |
| Central MA Housing Alliance Furniture Exchange (508) 791-7265 | 7-11<br>Bellevue | Worcester | MA | 01609 | |


**Supportive Services for Veterans and their Families:** VA aims to improve very low-income Veteran families' housing stability through the SSVF Program with outreach, case management, and assistance in obtaining benefits. Here is a list of SSVF Partners:

Lynn Housing Authority, Essex County & Middlesex County: 781-581-8640 Soldier On, Inc. /Berkshire, Hampshire, Franklin: 866-406-8449 Veterans Northeast Outreach Center Essex and Middlesex Counties, MA 978-372-3626 Veterans, Inc. /Worcester County: 800-482-2565 Vietnam Veterans Workshop, Inc. 617-371-1850 Vietnam Veterans Workshop, Inc./City of Boston (Suffolk County, only city)

Volunteers of America of Massachusetts, Inc./Suffolk, Middlesex, Plymouth, Norfolk,

Balance of State: 617-447-4287

617-371-1850


## Social Risk Factors Resource Guide: <u>LEGAL SUPPORT RESOURCES</u>

If you have any questions about the information provided below or want additional assistance contacting the programs, please contact Timothy Driscoll, 781-687-2374, Health Care for Homeless Veterans Program at Bedford VA.

#### Veteran Justice Outreach Program (VJO) 781-687-2377

VA Program providing support to VA eligible Veterans involved in the justice system. VJO Specialists provide direct outreach, assessment, case management, and pre-trial diversion through access to VA healthcare services.

**Center for Public Representation (413) 587-6265** [website will be provided here] Non-profit organization that provides legal assistance to consumers

#### Committee for Public Counsel Services (CPCS) (800) 882-2095

Provides free legal representation for consumers facing commitment hearings

#### Disability Law Center (800) 872-9992 [website will be provided here]

Non-profit organization that provides legal assistance for any person with a disability including consumers.

#### Mass. Correctional Legal Services (617) 482-2773

Non-profit advocacy organization for inmates

#### Mass. Law Reform Institute (617) 357-0700 [website will be provided here]

Non-profit agency that provides legal assistance, information and advocacy particularly for the poor and disenfranchised

#### Mass. Commission Against Discrimination (MCAD) (617) 727-3990

Assists in any discrimination case including workplace.

**Mental Health Legal Advisors Committee (800) 342-9092** [website will be provided here] Agency that provides legal assistance to consumers

#### Volunteer Lawyers Project (617) 423-0648

Network of attorneys that provide legal representation at reduced fees

#### Find Legal Help website [website will be provided here]

Features a state-by-state listing of legal help with links to basic legal information, lawyer referrals and free legal help. To find a pro bono program click on the "Free Legal Help" or "Pro bono".

#### Law Help website [website will be provided here]

Helps low- and moderate-income people find free legal aid programs in their communities as well as answers to questions about their legal rights.

**Pro Bono website** [website will be provided here]


Page **78** of **83** Version: 5/4/2021

A national, online resource for legal aid and pro bono attorneys, law professors and students, and related social services advocates.

VA Central IRB Effective Date: November 29, 2023

# Social Risk Factors Resource Guide: <u>EXPOSURE TO VIOLENCE AND/OR ABUSE RESOURCES</u>

If you have any questions about the information provided below or want additional assistance contacting the programs, please contact Timothy Driscoll, 781-687-2374, Health Care for Homeless Veterans Program at Bedford VA.

#### **Resources for Crisis/Emergency Response**

For immediate need, dial 911 or report to local emergency room/urgent care.

#### **Edith Nourse Rogers Memorial Veterans Hospital - VA Police**

Description: VA Campus Police at Edith Nourse Rogers Memorial Veterans Hospital (Bedford,

MA)

Contact: Emergency line: 781-687-2555. NON-Emergency line: 781-687-2404

Eligibility requirements: none

Cost: none

#### **Massachusetts Department of Children & Families**

**Description:** Massachusetts child abuse and neglect protection services **Contact:** Main line: 617-748-2000. Hotline to file report: 1-800-792-5200.

[website will be provided here]

Eligibility requirements: Legal minors under 18 and adults 18-22 transitioning out of DCF

care.

Cost: None

#### Massachusetts Department of Elder Services (person is over age 60)

**Description:** If a person over the age of 60 and living in the community experiences physical, sexual, or emotional abuse, caretaker neglect, financial exploitation, or self-neglect.

Contact: 1-800-922-2275. (If abuse by nursing home or hospital, contact Department of Public

Health at 1-800-462-5540). [website will be provided here]

Eligibility requirements: People over the age of 60 and living in the community.

Cost: None

#### **Massachusetts Disabled Persons Protection Commission**

**Description:** Protection of adults with disabilities from serious physical and/or emotional injury

from acts and/or omissions from their caregivers.

[website will be provided here] **Contact:** 1-800-426-9009

Eligibility requirements: Adults with disabilities.

Cost: None

#### Resources for Treatment/Clinical Care

#### **Mental Health Clinic Recovery Services**

**Description:** Outpatient mental health treatment with comprehensive behavioral health teams

(i.e., psychiatry, nursing, psychology, social work staff).

Contact: 781-687-2347


Eligibility requirements: Eligible for VA care.

Cost: Visit copay if applicable

**Safing Center** 

**Description:** Outpatient therapy focused on treatment and prevention of intimate partner

violence. [website will be provided here]

Contact: 781-687-3998

**Eligibility requirements:** Veteran eligible for VA care. Non-veteran collaterals (e.g., partners)

can receive couples therapy with the veteran or up to 4 individual therapy sessions.

Cost: Visit copay, if applicable.

Military Sexual Trauma (MST) Coordinator

**Description:** Resource for eligibility and treatment coordination related to sexual assault.

Contact: 781-687-3226

Eligibility requirements: Eligible for VA care.

**Cost:** Visit copay if applicable.


## Social Risk Factors Resource Guide: <u>EMPLOYMENT RESOURCES</u>

If you have any questions about the information provided below or want additional assistance contacting the programs, please contact Timothy Driscoll, 781-687-2374, Health Care for Homeless Veterans Program at Bedford VA or John Bowers, 781-687-2575, Vocational Rehab Specialists at Bedford VA.

#### **Veterans Employment Resources / Vocational Support**

Description: A variety of services to help veterans re-entering the workforce including

transitional work, supported employment and job search assistance

Contact: John Bowers / Paul Cheney 781-687-2575

Eligibility requirements: Eligible for VA Care; Determined by VA admissions

Cost: None

## Massachusetts Rehabilitation Commission ("Mass Rehab")

**Description:** The Vocational Rehabilitation Program helps people with disabilities get and keep

a job.

Contact: Main number: 617- 204-3600

Eligibility requirements: Have a disability. Want to work and need Vocational Rehabilitation

services to train, find, or keep a job.

Cost: None

#### Vocational Rehabilitation and Employment (VR&E)/Veterans Benefits Administration

**Description:** Vocational Rehabilitation and Employment (VR&E) services to help with job training, employment accommodations, resume development, and job seeking skills coaching **Contact:** [website will be provided here]

**Eligibility requirements:** Have a service connected disability of at least 10%. Have a discharge other than dishonorable.

Cost: None

\*\*Please note: Veterans Employment Resources also offers connection to pro bono legal services and child support assistance. Please contact Paul Cheney at 781-687-2575 for information on the legal clinic and Debra Locke at 781-687-2427 for information on the child support clinic.


#### Social Risk Factors Resource Guide: SOCIAL SUPPORT

If you have any questions about the information provided below or want additional assistance contacting the programs, please contact Anthony Russo, 781-687-3322 or [email available], Health Technician at Bedford VA.

#### **VA Community Recovery Connections Program**

**Description:** Information about Veteran peer support groups, community-based self-help groups, and other group-based opportunities to connect with other Veterans and civilians.

**Contact:** Tony Russo 781-687-3322

Eligibility requirements: Eligible for VA Care; Determined by VA admissions

Cost: None

#### **VA Social Skills Educational Opportunities**

**Description:** Education and training for Veterans interested in increasing their social skills and broaden their connections to Veterans and civilians around them. Services include individual and group trainings and coaching to build social support.

Contact: Michelle Esterberg 781-687-3935

Eligibility requirements: Eligible for VA Care; Determined by VA admissions

Cost: None

#### Name of program / resource: Veteran Coffee Socials

**Description:** Open weekly community-based meetings of Veterans in 22 communities in the local area. The only agenda is for Vets to get together to connect with other Vets, share information and support, and watch out for other Veterans in that community. These are free-standing independent groups.

**Contact:** Steven Hines (781-687-3173) can provide a listing of Veteran Coffee Socials time and location.

Eligibility requirements: None – open to all.

Cost: None


# Appendix P. Mail and Email Text for Delivering Resource Sheets to Veterans

#### 1. Cover Letter to Veterans mailed with Resource Sheets:

Veterans' Resource Needs Study (Address of Site location) (Phone number for Site RA)

(Date)

Hello, and thank you for participating in our study!

When we spoke on the phone several days ago, I promised to mail you some written material on agencies and programs that may be able to help you with the needs that you identified.

Please read through the enclosed material, and contact any of the listed programs or services directly at any time.

If you have questions about enclosed material, please call me at the number above.

Thank you.

#### 2. Email message to Veterans who choose to have Resource Sheet emailed:

Hello, and thank you for participating in our study!

The written material about Veterans' resources that I mentioned on the phone today is attached to this message for you to download and open. You will also receive a printed copy in the mail in a few days.

Thank you.

\*This email and attachment were sent with privacy encryption.

PLEASE DO NOT REPLY TO THIS MESSAGE. This is not a regularly maintained account and a response cannot be guaranteed. Should you need to connect with us, please call (insert site RA phone number).
